

# RESEARCH PROTOCOL

Final Version 1.0\_30<sup>th</sup>November 2021 Final Version 1.1\_10<sup>th</sup>December 2021 Final Version 1.2\_20<sup>th</sup>December 2021 Final Version 1.3\_19<sup>th</sup>January 2022 Final Version 1.4\_3<sup>rd</sup> March 2022 Final Version 1.5\_22<sup>nd</sup>. March 2022

# **Title**

Validation of Bulbicam for use on patient suffering from Diabetic retinopathy (DR) and Age-related macular degeneration (AMD)

**EudraCT number: 2021-006258-30** 

ClinicalTrial.gov: NCT

Protocol number: V1 OTH/DR; AMD-I/2022

# **Sponsor**

BulbiTech A/S, Dybdahls veg 5, Trondheim, Norway

# Administration

**Project Manager: Prof Stig Larsen** 

Responsible Ophthalmologist: Prof Goran Petrovski

Project Coordinator: Bård Dalhøi

#### CONFIDENTIAL

The information in this document is confidential and will not be disclosed to others without written authorization from Bulbitech A/S except to the extent necessary to obtain informed consent or for discussions with regulatory authorities, Independent Ethics Committees (IECs) or persons participating in the conduct of the study.

# **0:** Steering committee

The study will be administered by a steering committee headed by Prof Stig Larsen. The members of the committee are:

Project manager: Professor Emeritus Stig Larsen; Norwegian University of Life

Sciences / Meddoc AS, Hvamstubben 14 2013 Skjetten

Project coordinator: Bård Dalhøi. MSc Osteopathy

Chief Executive Officer (CEO) BulbiTech AS Trondheim

Responsible Ophthalmology: Professor Goran Petrovski Dr Med, MD, Ophthalmologist

Department of Ophthalmology, Oslo University Hospitals /

Ullevål Hospital, Oslo

PhD-fellow: Dr Bjørn Helland Hansen MD, Ophthalmologist

Department of Ophthalmology, Oslo University Hospitals /

Ullevål Hospital, Oslo

PhD-supervisors: Prof Goran Petrovski and Prof Emeritus Stig Larsen

The steering committee is responsible of:

1) The communication between the investigational sites

2) Supplementing study material to the sites

3) Continues data clarification

4) Corrections and amendments to the protocol

5) Publication of the results

BulbiCam; Validity study:

Other central participants in this study are:

Investigators: -Dr Alexander Sverstad MD, Ophthalmologist

Department of Ophthalmology, Oslo University Hospitals /

Ullevål Hospital, Oslo

-Dr Eivind Hovden Augustsen MD, Ophthalmologist Department of Ophthalmology Helgeland Sykehus

-Dr Henrik Skaret, Ophthalmologist

Department of Ophthalmology Helgeland Sykehus

Responsible statistician: Hans E Fagertun; MS Mathematical Statistics with specialty in

Biostatistics Meddoc A/S, Hvamstubben 14, 2013 Skjetten

Data Manager: Vivy Liang Larsen; MS, Data Manager Meddoc A/S,

Hvamstubben 14, 2013 Skjetten

Clinical Monitor: Sakaoduean Phonphimai; BS, CRA Meddoc A/S

Hvamstubben 14 2013 Skjetten

The study will follow the ethical guidelines for health-related research involving humans prepared by CIOMS and conducted in compliance with the protocol.<sup>1</sup>

Prof Stig Larsen has written the trial protocol and is responsible for writing the clinical study report (CSR) with supports and corrections from the steering committee and the participating investigators. Hans E Fagertun is responsible for the statistical analysis supported by Stig Larsen. The data management and the clinical monitoring will be headed by Vivy Liang Larsen supported by members from the clinical- and the DM-group.

The result shall be published in an international medical journal and the manuscript prepared by the steering committee and the investigator. All participating centers shall be represented in the list of authors.

# 0.1: Signature Sheet

#### Protocol Authorized:

Stig Larsen<sup>1</sup>, Goran Petrovski <sup>2</sup>, Bjørn Helland Hansen<sup>3</sup> and Bård Dalhøi<sup>4</sup>

# Qualifications:

- 1. Project Manager, Professor; Controlled Clinical Trials Research Methodology and **Biostatistics**
- 2. Professor; Ophthalmology
- 3. PhD-fellow; Ophthalmology
- 4. Project Coordinator, CEO BulbiTech A/S

| Signature 1 | Date |
|-------------|--------|
| Signature 2 | . Date |
| Signature 3 | . Date |
| Signature 4 | Date |

#### 0.2: Contact names and addresses

Professor Stig Larsen; Clinical Research Methodology and Statistics

Project Manager, Norwegian University of Life Sciences / Meddoc A/S, Hvamstubben 14,

2013 Skjetten

Phone +47 413 26 325 E-mail: sl@meddoc.no

Professor Goran Petrovski; Ophthalmology

Department of Ophthalmology, Oslo University Hospitals / Ullevål Hospital, Oslo

Phone: +47 9222 6158

E-mail: goran.petrovski@medisin.uio.no

Dr Bjørn Helland Hansen

Chief Medical Officer (CMO)

BulbiTech AS, Dybdahlsveg 3 – 5, 7051 Trondheim

Phone: +47 412 35 584 E-mail: bjorn@bulbitech.com

Bård Dalhøi CEO BulbiTech AS

**Project Coordinator** 

BulbiTech AS, Dybdahlsveg 3 – 5, 7051 Trondheim

Phone: +47 90 99 01 99 E-mail: bard@bulbitech.com

Dr Alexander Sverstad MD, Ophthalmologist

Department of Ophthalmology, Oslo University Hospitals / Ullevål Hospital, Oslo

Phone: +47 9946 1682

E-mail: <u>alexsvers@gmail.com</u>

Dr Henrik Skaret, Ophthalmologist

Department of Ophthalmology Helgeland Sykehus

Phone: +47 46446640

E-mail: <u>henrik.skaret@gmail.com</u>

Vivy L Larsen MSc Data Manager (DM)

Meddoc AS, Hvamstubben 14, 2013 Skjetten

Phone: +47 412 93 161 E-mail: vll@meddoc.no

Hans E Fagertun MS

Statistician

Meddoc AS, Hvamstubben 14, 2013 Skjetten

Phone: +47 412 93 161 E-mail: hf@meddoc.no

Einar Kvam Lundberg BS Data engineer/programmer

Meddoc AS, Hvamstubben 14, 2013 Skjetten

Phone: +47 951 79 012 E-mail: ekl@meddoc.no

# 0.3: List of Abbreviations

| Abbreviation | Explanation |
|--------------|-------------------------------------------------------------|
| AE | Adverse Event |
| AMD | Age related macular degeneration |
| BCAM | Bulbicam |
| BSC | Bachelor of Science |
| EMP | Eye Movement Perimeter |
| CIOMS | Council for International Organizations of Medical Sciences |
| CSR | Clinical Study Report |
| CRD | Clinically Relevant Difference |
| CRF | Case Report Form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CV | Curriculum Vita |
| DA | Dark adaptation |
| DR | Diabetes retropathy |
| DM | Data Management |
| DME | Diabetic macular edema |
| EQ-5D-5L | QoL questionnaire |
| GCP | Good Clinical Practice |
| HC | Healthy Control |
| ITT | Intention to treat |
| LOCS | Lens Opacification classification system |
| LOCF | Last Observation Carried Forward |
| MSC | Master of Science |
| NPDR | non-proliferative stage |
| NSD | Norwegian Centre for Research data |
| OTH | Ophthalmology |
| OR | Odds Ratio |
| PCIOL | Posterior Chamber Artificial Ocular Lens |
| PDR | proliferative stage |
| PP | Per Protocol |
| PhNR | Photonic negative response |
| PDR | Proliferative DR |
| PIPR | Post-illumination pupil response |
| PSC | Posterior Sub Capsular |
| QoL | Quality of Life Questionnaire |
| RAPD | Relative Afferent Pupil Defect |
| REK | Regional Ethical Committee |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis System |
| SD | Standard Deviation |
| SFT | Swinging flashlight test |
| ST | Standard Method |
| SOC | System Organ Class |
| SURSAR | Suspected Unexpected Serious Adverse Reactions |
| VAS | Visual Analogue Scale |
| 7 1 10 | 1 10001 1 111010500 Douto |

# 0.4: Distribution of Clinical trial Protocols

| Complete Version | Date | Writer | Receivers | Internal | Date released |
|---|---|---|---|---|---|
| | | | | review | |
| Version 0.1 | 28.10.2021 | SL | BD, GP, BHH, HF, VL, EL | Yes | No |
| Version 0.2 | 02.11.2021 | SL | BD, GP, BHH, HF, VL, EL | Yes | No |
| Version 0.3 | 15.11.2021 | SL | BD, GP, BHH, HF, VL, EL, AS, HS | Yes | No |
| Final Version 1.0 | 30.11.2021 | SL | BD, GP, BHH, HF, VL, EL, AS, HS | No | 30.11.2021 |
| Final Version 1.1 | 10.12.2021 | SL | BD, GP, BHH, HF, VL, EL, AS, HS | No | 30.11.2021 |
| Final Version 1.2 | 20.12.2021 | SL | BD, GP, BHH, HF, VL, EL, AS, HS | No | 30.11.2021 |
| Final Version 1.3 | 19.01.2022 | SL | BD, GP, BHH, HF, VL, EL, AS, HS | No | 30.11.2021 |
| Final Version 1.4 | 03.03.2022 | SL | BD, GP, BHH, HF, VL, EL, AS, HS | No | 03.03.2022 |
| Final Version 1.5 | 22.03.2022 | SL/BHH | BD, GP, HF, VL, EL, AS, HS | No | 03.03.2022 |

SL: Stig Larsen BD: Bård Dalhøi GP: Goran Petrovski

BHH: Bjørn Helland Hansen

HF: Hans Fagertun VL: Vivy Larsen EL: Einar Lundberg AS: Alexander Sverstad HS: Henrik Skaret

# 0.5: Participating Institutions

BulbiCam; Validity study:

The study will be performed as a multicenter study at Oslo University Hospitals/Ullevål and Helgeland Hospital.

# Content

| 0: Steering committee | 1 |
|-------------------------------------------------------------------|----|
| 0.1: Signature Sheet | |
| 0.2: Contact names and addresses | |
| 0.3: List of Abbreviations | 5 |
| 0.4: Distribution of Clinical trial Protocols | 6 |
| 0.5: Participating Institutions | |
| I: Protocol Synopsis | |
| 1.1: Title | |
| 1.2: Protocol number | 10 |
| 1.3: Aim | |
| 1.4: Study population | |
| 1.5: Trial equipment | |
| 1.6: Design | |
| 1.7: Variables | |
| 1.7.1 Main Variables | 11 |
| 1.7.2 Supporting Variables | |
| 1.8: Study procedure | |
| 1.9: Sample size | |
| 1.10: Time schedule | 13 |
| 1.11: Flow chart | 13 |
| II: Introduction | |
| 2.1: Background | |
| 2.1.1:Diabetic Retinopathy (DR) | |
| 2.1.2: Age-related macular degeneration (AMD) | |
| 2.2: BulbiCam | |
| 2.4: Objective | |
| III: Population and sampling | |
| 3.1: Reference population | |
| 3.2.1: Inclusion criteria; study population 1 (DR) | |
| 3.2.2: Exclusion criteria; study population 1 (DR) | |
| 3.2.3: Inclusion criteria; study population 2 (AMD). | |
| 3.2.4: Exclusion criteria; study population 2 (AMD) | |
| 3.2.5: Inclusion criteria; study population 3 (HC) | |
| 3.2.6: Exclusion criteria; study population 3 (HC) | |
| 3.3: Recruitment of patients | |
| 3.4: Benefit and risk assessment | |
| IV: Design | |
| 4.2: Stratification | |
| 4.3: Identification of patients | |
| <b>V: Evaluation</b> 5.1: Main variables | |
| 5.1.1: BulbiCam investigation | |
| 5.2: Secondary variables | |
| 5.2.1: Quality-of- Life questionnaires <sup>30</sup> | 23 |
| 5.2.2: Common Terminology Criteria for Adverse Events version 4.0 | 25 |
| 5.3: Patient factors | |
| VI: Study procedure | |
| 6.1: Trial equipment and clinical procedure | 29 |

| 6.2: Inclusion visit and Screening phase | 29 |
|--------------------------------------------------------|----|
| 6.3: Study procedure | |
| 6.3.1: Part one (Repeatability) | 29 |
| 6.3.2: Part 2 (Stability) | |
| 6.4: End of the study | |
| 6.5: Stopping rule | 30 |
| 6.6: Report of serious adverse effect (SAE) | 30 |
| 6.7: Study duration | 30 |
| VII: Project management and Monitoring | 31 |
| 7.1: Project management | 31 |
| 7.2: Publication of the results | 31 |
| 7.3: Quality assurance demands | 31 |
| 7.4: Start-up and closing visit | |
| 7.5: Monitoring procedure | |
| 7.6: Curriculum vitae | |
| 7.7: Site file | |
| VIII: Data Management | |
| 8.1. Case Record Forms (CRF) | |
| 8.2. Study Database | |
| IX: Discontinuation | |
| 9.1: Discontinuation not related to the study question | |
| 9.2: Discontinuation related to the study question | |
| X: Ethical consideration | |
| 10.1: Consideration of steering committee | |
| 10.2: Approval of the project | |
| 10.3: Informed consent | |
| 10.4: Protection of personal data | |
| XI: Statistical model | |
| 11.1: Handling of discontinuation | |
| 11.2: Presentation of the result | |
| 11.3: Sample size | |
| XII: Operational matters | |
| 12.1: Investigator's agreement | |
| 12.2: Instructions | |
| 12.3: Amendments to the protocol | |
| 12.4: Protocol deviations | |
| 12.5: Compliance monitoring | |
| 12.6: Responsibilities | |
| 12.7: Confidentiality | |
| 12.8: Investigator and Sponsor withdrawals | |
| XIII: References | |
| XIV: Amendments | 42 |
| XV: Appendix | 45 |
| 15.1: Set of CRF's | |
| 15.1.1: CRF I; Inclusion and exclusion | 45 |
| 15.1.2: CRF II; Demographic factors | |
| 15.1.3: CRF III; Medical history | |
| 15.1.4: CRF IV; Quality of life | |
| 15.1.6: CRF VI; Adverse Events | |
| 15.1.7: CRF VII; End of Trial | |
| 15.2: Bulbicam Certificate | |

| 15.2.1: ISO-Certificate | 55 |
|-----------------------------------------------------|----|
| 15.2.2: Certificate of free Sales | 56 |
| 15.3: CV; Primary investigator & Steering Committee | |
| 15.3.1: Bård Dalhøi CEO BulbiTech AS | |
| 15.3.2: Professor Goran Petrovski; Ophthalmology | 60 |
| 15.3.3: Professor Stig Larsen | |

# I: Protocol Synopsis

#### 1.1: Title.

Validation of Bulbicam for use on patient suffering from Diabetic retinopathy ((DR) and Agerelated macular degeneration (AMD)

#### 1.2: Protocol number

Protocol number: V1 OTH/DR; AMD - I/2022

#### 1.3: Aim

- To investigate repeatability and stability of the six OTH-related Bulbicam tests in patients suffering from a) Diabetic retinopathy (DR), b) Age related macular degeneration (AMD) and matched healthy controls (HC).
- To compare Bulbicam and the Standard Method on measurements of Visual Field and Pupil
- To contribute to the establishment of normal range for DR and AMD patients with different degree in the disease development related to the Bulbicam tests.
- To contribute to the establishment of normal range for a normal population without eye-disease related to the Bulbicam tests.

# 1.4: Study population

The study consists of the following three study populations: 1) Patients suffering from DR of both genders above 18 years of age with different disease degree; 2) Patients suffering from AMD of both genders above 18 years of age with different disease degree; 3) Gender- and age-matched HC without any eye diseases.

#### 1.5: Trial equipment

Bulbicam will be used in the study and the following six tests will be performed at each investigation: "Neurofield 64", "Ptosis", "Dynamic Acuity", "Dynamic Contrast ", "Dark Adoption" and Pupil. The Standard Method will be used initially for measurements of "Neurofield64", "Visual Field" and "pupil".

# 1.6: Design

The study will be performed as a controlled, open, and non-randomized, stratified observational multicenter study. The stratification factors are the pathology of DR and AMD and the degree of disease. Within each of the four strata, healthy matched controls related to gender- and age (1:1) will be included. The degree of DR is defined as follows:

- 1) Mild retinopathy: Mild nonproliferative diabetic retinopathy
- 2) Moderate retinopathy: Moderate nonproliferative diabetic retinopathy The degree of AMD is defined as follows:
  - 1) Early AMD
  - 2) Intermediate

For each included patient, a gender- and age-matched HC will be included. All included participants will perform Bulbicam eye-investigation twice at three flowing days with a rest period of at least one hour. Each investigation includes same six Bulbicam tests. The Standard method will only be performed once as the first investigation at day 1 for measurements of "Visual Field" and Pupil"

# 1.7: Variables

#### 1.7.1 Main Variables

BulbiCam; Validity study:

The main variables will be the variables recorded at the six Bulbicam tests described in the table below:

| TEST | VARIABLE | UNIT | FORMAT |
|---|---|---|---|
| | Seen/unseen (0) | 0= unseen target | xml. |
| | Saccadic Reaction Time | Ms - 4 digits, 0 decimals | xml. |
| Visual Field | Angular deviation | Degree - 3 digits, 0 decimals | xml. |
| | X-coordinate | Degree - 2 digits, 0 decimals | |
| | Y-coordinate | Degree - 2 digits, 0 decimals | |
| Ptosis | MDR1 | mm - 2 digits, 2 decimals | xml. |
| 1 10515 | MDR2 | mm - 2 digits, 2 decimals | xml. |
| Dynamic Acuity | Visual acuity | LogMAR 1 digit, 2 decimals | xml. |
| Dynamic Contrast | Contrast sensitivity | ConRatio 1 digit, 2 decimals | xml. |
| Dark Adaptation | Fixed contrast | Hz 1 digit, 1 decimal | xml. |
| Dark Adaptation | Fixed frequency | ConRatio 1 digit, 2 decimals | xml. |
| | Diameter (mm) | mm - 1 digit, 2 decimals | xml. |
| Pupil | Peak velocity | mm/s - 1 digit, 2 decimals | xml. |
| | Latency | Ms - 3 digits, 0 decimals | xml. |
| | RAPDlog | 1 digit, 2 decimals | xml. |

LogCon defined as  $-\log 10$  (contrast ratio), EG if the low brightness part of the stimulus is 2 nits, the high brightness part 255 nits, the LogCon would be  $-\log 10$  (2/255) =2, 1.

# 1.7.2 Supporting Variables

The supporting variables will be recorded by the Standard (ST) investigation for DR and AMD.

| Test | No of instances | Variable | Unit | Unit description |
|---|---|---|---|---|
| GAT | 1 | Pressure | mmHg | 2 digits, 1 decimal |
| iCare | 1 | Pressure | mmHg | 2 digits, 1 decimal |
| Acuity chart | 1 | Visual acuity | logMAR | 1 digit, 1 decimal |
| Contrast chart | 1 | Contrast acuity | Pelli-Robson score | 1 digit, 2 decimals |
| | 1 | Nasal step | | |
| | 1 | Temporal wedge | | |
| | 1 | Partial arcuate (sup) | | |
| | 1 | Partial arcuate (inf) | | Boolean |
| | 1 | Arcuate (sup) | Present | (true / false) |
| | 1 | Arcuate (inf) | | (true / faise) |
| | 1 | Altitudinal (inf) | | |
| | 1 | Altitudinal (sup) | | |
| | 1 | Paracentral | | |
| | | MD | dB | 2 digits, 2 decimals |
| Visual field | 54 | X coordinate | Degrees | 3 digits, 1 decimal |
| | | Y coordinate | Degrees | 3 digits, 1 decimal |
| | 1 | Threshold sensitivity | dB | 2 digits, 2 decimals |
| | 1 | Percentile degree | Score 1-5 | 1 digit |
| | 1 | Defuse defect | dB | 2 digits, 1 decimal |
| | 1 | Local defect | dB | 2 digits, 1 decimal |
| | 1 | sLV | dB | 2 digits, 1 decimal |
| | 1 | False positive | Percent (Reliability) | 2 digits |
| | 1 | False negative | Percent (Reliability) | 2 digits |
| | 1 | Reliability factor | Percent (Reliability) | 2digits, 1 decimal |
| | 1 | Mean Sensitivity | dB | 2 digits, 1 decimal |
| OCT RNFL | 1 | Average thickness | μm | 3 decimals |
| OCT GCL | 1 | Volume | mm^3 | 3 decimals |
| Pupil | 1 | Diameter change (max-min) | mm | 1 digit, 2 decimals |

The central variables related to DR and AMD will be "RAPD NDF", "Seen /unseen "," Time until the given point is recorded as seen", "the light in decibel when the point is seen", X- and Y-coordinates and "Pupil diameter in mm" and "OCT RNFL".

#### 1.8: Study procedure

BulbiCam; Validity study:

Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will receive an appointment for starting the study. The Bulbicam examination will be performed twice a day with a rest period of one hour between each registration. This procedure will be repeated the following two days. All demographic data, social factors and history of disease will be recorded at screening. Additionally, the quality of life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded initially as individual baseline values.

The Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be used for measuring and classifying the tolerability and toxicity at the end of each day of investigation.

# 1.9: Sample size

Sixteen DR patients and 16 AMD patients from each of the two categories will be recruited from the two participating hospitals. All together a total of 16x2=32 patients will be included. For each included patient, one gender- and age-matched HC will be recruited. In total 32 HC.

#### 1.10: Time schedule

The study duration for each participant will be 3 days including six measurements using Bulbicam and one using the Standard method. The recruitment period is nine months. The total duration of the study will be as follows:

| Inclusion of the first patient with control | 01-05-2022 |
|---------------------------------------------|------------|
| End of trial; last patient with control | 15-01-2023 |
| Closing database | 15-02-2023 |
| Finalized Clinical Study Report | 01-03-2023 |

#### 1.11: Flow chart

| | Screening | Day 1; | Day 2; | Day 3; |
|---|---|---|---|---|
| | | Repeatability | Stability-1 | Stability-2 |
| Inclusion and Exclusion criteria | X | | | |
| Oral & written informed consent | X | | | |
| Patient factors | X | | | |
| History of disease | X | | | |
| Eye-examination. | X | | | |
| Concom. Medicine | X | X | X | X |
| Quality of Life | X | | | |
| | Bulbica | am tests | | |
| Visual Field | | X | X | X |
| Ptosis | | X | X | X |
| Dynamic Acuity | | X | X | X |
| Dynamic Contrast | | X | X | X |
| Dark Adaption | | X | X | X |
| Pupil | | X | X | X |
| | Standard | d Method | | |
| GAT | | X | | |
| ICare | | X | | |
| Visual Field | | X | | |
| Pupil | | X | | |
| OCT RNFL | | X | | |
| OCT GCL | | X | | |
| Adverse Events [CTCAE] | X | X | X | X |
| End of study | | | | X |

# **II: Introduction**

#### 2.1: Background

BulbiCam; Validity study:

2.1.1:Diabetic Retinopathy (DR) remains a common complication of diabetes mellitus and is a leading cause of vision loss elderly population globally. Among those with diabetes, global prevalence was 22.27% (95% confidence interval, 19.73-25.03%) for Diabetic retinopathy, 6.17% (95% CI 5.43-6.98%) for vision-threatening DR and 4.07% (95% CI 3.42-4.82%) for clinically significant macular edema.<sup>3</sup> The prevalence of DR in Indian population with DM was 19% (95% CI 16-20.1%).4 DR prevalence was highest in Africa (35.90%), and North American and Caribbean regions (33.30%); and lowest in South and Central America region (13.37%). In meta-regression models adjusting for habitation type, response rate, study year and DR diagnostic method, Hispanics (odds ratio [OR], 2.92; 95% CI, 1.22-6.98) and Middle Easterners (OR, 2.44; 95% CI, 1.51-3.94) with diabetes were more likely to have DR, compared to Asians.<sup>2</sup> The major risk factors of DR include disease duration, poor glycaemic control, presence of hypertension, higher body mass index, puberty, pregnancy, and cataract surgery. Early detection and treatment can prevent any diabetic-related visual impairment. To reduce the impact of DR-related visual loss, it is important to look for innovative ways of managing and preventing diabetes and optimize cost-effective screening programs within the community.

Diabetic Retinopathy can be clinically characterised into a non-proliferative (NPDR) stage and proliferative (PDR) stage depending on the retinal vascular lesions. It can also lead to fluid accumulation in the retina called diabetic macular edema (DME). Visual functions are affected in the early and late stage of the disease. Current research shows that contrast sensitivity is a more sensitive tool to detect early retinal changes than visual acuity. In a recent study contrast sensitivity score was noted to be significantly lower in diabetic patients with no retinopathy and mild nonproliferative retinopathy. 5 Cone photoreceptor light sensitivity is responsible for light adaptation and rod light sensitivity for dark adaptation and performance. Studies on retinal neurodegeneration in DM have reported abnormalities of inner-retina structure and function. These include reduced retinal ganglion cell thickness, abnormal ERG patterns i.e., reduced photonic and scotopic response. Delay in high-frequency flicker ERG and reduced cone sensitivity have been reported in early cases that can serve as a screening tool. Reduction in pattern ERG, photonic negative response (PhNR) and the postillumination pupil response (PIPR) have been reported in diabetic patients with and without NPDR. Light and dark adapted steady state pupil size and melanosis mediated pupil light reflex are reduced in diabetes and all stages of DR. 8,9 These proof-of-concept studies demonstrate that chromatic pupilometer methods can serve as a screening and early detection tool to assess the damage to photoreceptors of retinal/optic nerve diseases. Dark adaptation is being reported to be affected in retinal dysfunction conditions such as ARMD, Diabetic Retinopathy and Retinitis Pigmentosa. In addition to the effect of early DR on cone-mediated light sensitivity, the second most impaired visual function was rod-mediated visual sensitivity. These indicate diabetes exerts early impact on the inner and outer retinal function. 10 Dark adaptation was measured in NPDR using AdaptDx dark adaptometer (MacuLogix, IncHummelstown, PA, USA) and the results suggested that RPE and photoreceptor cell dysfunction was noted to be progressed with worsening DR and rod recovery dysfunction occurred earlier than cone dysfunction.<sup>11</sup>

2.1.2: Age-related macular degeneration (AMD) is the main cause of adult blindness in the Western world. The prevalence of advanced AMD in two studies were 1,6% and 1,5% respectively, and the incidence of AMD in the population of >75 years of age is significantly

growing, which is becoming a big public health problem as the population of elderly is expected to increase by 54% between 2005 and 2025 in a Western population <sup>12,13</sup>.

In developing countries there is little data on the prevalence of the disease<sup>3</sup>.

In a study from India, there is evidence that AMD may exist to the same extent as it does in developed countries. The prevalence of early (dry form) and late (wet form) stages of AMD is like that observed in Western populations. The prevalence in the age of >80 years seems to be underestimated <sup>14</sup>. In countries with growing elderly populations, it is important for society to plan for low-vision services and rehabilitation, which implies the need for early detection of AMD.

Research states subjects in the early stages of dry AMD have delayed dark adaptation (DA), which indicates a delay of light sensitivity by the photoreceptors (cones and rods), which have been exposed to bright light 15-21. The photoreceptors of cones and rods are slowly increasing their sensitivity to light in a dim environment. Cones adapt faster, so the first few minutes of adaptation is related to the cone moderated vision. Rods adapt slower, but can adapt to dimmer illuminations, and they replace the cone mediated period. The method of functionally assessing DA in early detection of dry AMD is described in multiple studies. Patients with dry AMD have problems with their vision under low light conditions. Therefore, the functional sign of early AMD is the lack of the subject's ability to adapt in the dark after being exposed to light. The rod photoreceptor cells are extremely sensitive and can be triggered by a single photon <sup>22-23</sup>. Cone photoreceptor cells improve sensitivity quickly and recover their total function after 5 to 10 minutes. There is a transition from cone to rod function in dark adaptation, and the rod responses to changes in light level is thought to be slow as the rods take 20 to 40 min to fully recover after the offset of a bright light <sup>24</sup>. Although rod recovery is affected in early AMD, cone sensitivity is investigated also to be an effective index of early AMD detection<sup>25-26</sup>. To clinically investigate the rod adaptation is time consuming for the patient and may last up to 20 to 40 minutes, whereas cone adaptation should not take longer than 1-2 minutes, as cones take up to 2 min to recover in the dark. As both cones and rods are affected in early AMD, it is more time saving to investigate the cone DA effort.

When bleaching the retinal photo pigments exposed to lower light levels, there is an adaptation in the retinal neurons fed by the cones. The approximate time for recovery in the dark after moderate light adaptation is said to be  $\pm$  15 sec in the blue/yellow pathway<sup>27</sup> and  $\pm$  20 s in the red/green pathway for the recovery<sup>28</sup>. It is even shown that there is a very rapid adaptation that takes less than 0.6 sec<sup>29</sup>. AMD usually classifies as "Early" and "Intermediate".

#### 2.2: BulbiCam

BulbiTech AS has developed a hardware/software product combination to simplify neuro-ophthalmic examinations. The multi-test device, BulbiCam (BCAM), is a combined eye tracking; pupil metric; video graphic dual device which include the following 10 tests under development and ready for validation:

- 1. 26 grids glaucoma screening perimetry
- 2. 64 grids full perimetry (NeuroField64)
- 3. Pupil and Relative Afferent Pupil Defect (RAPD) assessment
- 4. Semi-automatic ptosis (droopy eyelid) grading
- 5. Video-based nystagmus test
- 6. Dynamic acuity and contrast sensitivity test
- 7. Dark adaptation test
- 8. Smooth pursuit eye movements
- 9. Saccade movements

#### 10. Eye fixation stability

BCAM is connected to the BulbiHub software where measured data is stored and presented in numbers, diagrams, and graphs.

#### 2.3: Standard Method

Standard Method (ST) is the notation used for the golden eye-examination standard today. The supporting variables will be recorded by the Standard (ST) investigation for DR and AMD.

Table 1: Standard examination

| Test | No of instances | Variable | Unit | Unit description |
|---|---|---|---|---|
| GAT | 1 | Pressure | mmHg | 2 digits, 1 decimal |
| iCare | 1 | Pressure | mmHg | 2 digits, 1 decimal |
| Acuity chart | 1 | Visual acuity | logMAR | 1 digit, 1 decimal |
| Contrast chart | 1 | Contrast acuity | Pelli-Robson score | 1 digit, 2 decimals |
| | 1 | Nasal step | | |
| | 1 | Temporal wedge | | |
| | 1 | Partial arcuate (sup) | | |
| | 1 | Partial arcuate (inf) | | Boolean |
| | 1 | Arcuate (sup) | Present | (true / false) |
| | 1 | Arcuate (inf) | | (true / faise) |
| | 1 | Altitudinal (inf) | | |
| | 1 | Altitudinal (sup) | | |
| | 1 | Paracentral | | |
| | | MD | dB | 2 digits, 2 decimals |
| Visual field | 54 | X coordinate | Degrees | 3 digits, 1 decimal |
| | | Y coordinate | Degrees | 3 digits, 1 decimal |
| | 1 | Threshold sensitivity | dB | 2 digits, 2 decimals |
| | 1 | Percentile degree | Score 1-5 | 1 digit |
| | 1 | Defuse defect | dB | 2 digits, 1 decimal |
| | 1 | Local defect | dB | 2 digits, 1 decimal |
| | 1 | sLV | dB | 2 digits, 1 decimal |
| | 1 | False positive | Percent (Reliability) | 2 digits |
| | 1 | False negative | Percent (Reliability) | 2 digits |
| | 1 | Reliability factor | Percent (Reliability) | 2digits, 1 decimal |
| | 1 | Mean Sensitivity | dB | 2 digits, 1 decimal |
| OCT RNFL | 1 | Average thickness | μm | 3 decimals |
| OCT GCL | 1 | Volume | mm^3 | 3 decimals |
| Pupil | 1 | Diameter change (max-min) | mm | 1 digit, 2 decimals |

# 2.4: Objective

BulbiCam; Validity study:

The objective in this study is to validate the six of the BCAM tests to be used in examination of patients suffering from DR or AMD. The specific aims of the study are:

- To investigate repeatability and stability of the six OTH-related BCAM tests in patients suffering from a) DR, b) AMD and c) gender- and age-matched HC.
- To compare BCAM and the Standard Method on measurements of Visual Field and Pupil to ensure that BCAM measures what is assumed to measure.
- To contribute to the establishment of normal range for DR and AMD patients with different degree in the disease development related to the BCAM tests.



# III: Population and sampling

# 3.1: Reference population

The reference population consists of patients either suffering from DR or AMD without other eye diseases.

#### 3.2: Study populations

#### 3.2.1: Inclusion criteria; study population 1 (DR)

Consists of patients diagnosed with DR of both gender; passed the age of 18 years; without any other eye disease; suffering from other know serious disease but have a health situation in accordance with expectations related to the age.

#### 3.2.2: Exclusion criteria; study population 1 (DR)

Patients fulfil at least one of the following criteria will be excluded from participation in the study:

- Other visual disturbances and blindness
- Posterior Chamber Intra Ocular Lens (PCIOL)
- Physical or psychiatric disease, which may disturb the measuring procedure
- Patients who are not able to perform eye movements, so no full paresis of any ocular muscles.
- Patients whose visual acuity is less more than 1 logMAR in any eye, as these will not be able to focus on the test stimuli.
- Patients whose visible part of the eye is abnormal, such as subconjunctival hemorrhages or deformed pupils.
- Patients whose pupils are not able to respond normally to dilation or contraction due to damaged nerves, mechanical damage of the pupil etc.
- Participating in another clinical trial with pharmaceuticals the last six weeks before start of this trial treatment.
- With known alcoholic and drug dependency
- Not able to understand information.
- Not willing to give written consent to participate in the study.

#### 3.2.3: Inclusion criteria; study population 2 (AMD)

Consists of patients diagnosed with AMD of both gender; passed the age of 18 years; without any other eye disease; suffering from other know serious disease but have a health situation in accordance with expectations related to the age.

# 3.2.4: Exclusion criteria; study population 2 (AMD)

Patients fulfilling at least one of the following criteria will be excluded from participation in the study:

- Other visual disturbances and blindness
- Posterior Chamber Artificial Ocular Lens (PCIOL)
- Physical or psychiatric disease, which may disturb the measuring procedure

- Patients who are not able to perform eye movements, e.g., full paresis of any ocular muscles
- Patients with visual acuity more than 1 logMAR, as they will not be able to focus on the test stimuli
- Patients whose visible part of the eye is abnormal, such as subconjunctival haemorrhages or deformed pupils.
- Patients whose pupils are not able to respond normally to dilation or contraction due to damaged nerves, mechanical damage of the pupil etc.
- With known alcoholic and drug dependency
- Not able to understand information.
- Not willing to give written consent to participate in the study.

#### 3.2.5: Inclusion criteria; study population 3 (HC)

The study population 3 consists of gender- and age-matched controls to patients in study population 1 or 2; passed the age of 18 years without any eye diseases; not suffering from other know serious disease and have a health situation in accordance with expectations related to the age.

# 3.2.6: Exclusion criteria; study population 3 (HC)

Patients fulfilling at least one of the exclusion criteria listed under either paragraph 3.2.2 or 3.2.4 will be excluded from participation in the study

#### 3.3: Recruitment of patients

The patients will be recruited from Oslo University hospital, Ullevål and Helgeland hospital. If necessary, private Ophthalmology clinics in Oslo will be asked for recruitment. All the investigations in the study will be performed by the same Ophthalmologist at the given hospital. The investigator informs the patients about the study, handing and collecting the written informed consent form. In case the patient fulfils the inclusion/exclusion criteria and willing to sign the consent form, the patient is included in the study. No data from possible participants included in the screening phase but not fulfils the inclusion/exclusion criteria will be recorded in the database. The included patient will be asked if he/she know any person with same gender and age; in good health condition without any eye disease which may participate as a control in the study. The potential controls will be contacted by the responsible investigator, obtain information about the study, and expected tasks. Controls willing to sign the consent form is included in the study. In case of lack in controls, requests among the hospital staff will be performed.

#### 3.4: Benefit and risk assessment

BulbiCam; Validity study:

BulbiCam is new equipment specially developed for clinical investigation of eye. It will simplify neuro-ophthalmic examinations; increase the quality- and benefit of the examinations; detecting earlier correct diagnoses and increase the knowledge of the disease development under treatment. BCAM do not harm neither to the patients nor to the investigator.

# IV: Design

#### 4.1: Study design

The study will be performed as a controlled, open and non-randomized, stratified observational multicenter. The two stratification factors will be ophthalmological diagnose and the severity of the disease.



Figure 1: The overall study design. The numbers 1 to 6 indicate the sequence of Bulbicam measurements and \*) the measurements using the Standard Method

#### 4.2: Stratification

The two main strata are DR and AMD. The patients within each of these two strata will be divided in two sub-strata depending on the disease severity. Within each of the main strata, a third stratum will consist of gender- and age-matched HCs to the patients included in the two other sub-strata.

The three sub-strata within DR will be:

- 1. Healthy gender- and age-matched controls
- 2. Mild retinopathy: Mild nonproliferative retinopathy
- 3. Moderate retinopathy: Moderate nonproliferative retinopathy

The three sub-strata within AMD will be:

- 1. Healthy gender- and age-matched controls
- 2. Early AMD
- 3. Intermediate AMD

#### 4.3: Identification of patients

All information in the database will be anonymized and the activation key is stored by the clinically responsible ophthalmologist. The patients will be given one study identification number of six digits. The Id-number is divided in two parts in which the first part consists of four digits based on; country; site; disease and degree of the disease. Within these four-digit groups, two digits running number will be created by the DB-system.

**Digit 1:** Indicate the country [1=Norway; 2=India i.e.]

Digit 2: Indicate hospital site [1 = Site 1/Ullevål; 2= Site 2/Helgeland i.e.]
 Digit 3: Disease [0= Control; 1=Gla; 2=Cat; 3=DR; 4=AMD; 5=MS, i.e.].
 Digit 4: Degree of disease [0= none; 1= Mild/Early; 2=Moderate/Intermediate;

3=Severe].

**Digit 5&6:** Running number within group [01= Patient 1; 02=Patient 2 i.e.]

#### V: Evaluation

#### 5.1: Main variables

#### 5.1.1: BulbiCam investigation

The main variables will be the variables recorded at the six Bulbicam tests described in the table below:

Table 2: The main variables with unit of the six Bulbicam test included in the study

| TEST | VARIABLE | UNIT | FORMAT |
|---|---|---|---|
| | Seen/unseen (0) | 0= unseen target | xml. |
| NeuroField64 | Saccadic Reaction Time | Ms - 4 digits, 0 decimals | xml. |
| | Angular deviation | degree - 3 digits, 0 decimals | xml. |
| Ptosis | MDR1 | mm - 2 digits, 2 decimals | xml. |
| 1 10515 | MDR2 | mm - 2 digits, 2 decimals | xml. |
| Dynamic Acuity | Visual acuity | LogMAR 1 digit, 2 decimals | xml. |
| Dynamic Contrast | Contrast sensitivity | ConRatio 1 digit, 2 decimals | xml. |
| Dark Adaptation | Fixed contrast | Hz 1 digit, 1 decimal | xml. |
| Dark Adaptation | Fixed frequency | ConRatio 1 digit, 2 decimals | xml. |
| | Diameter (mm) | mm - 1 digit, 2 decimals | xml. |
| Pupil | Peak velocity | mm/s - 1 digit, 2 decimals | xml. |
| | Latency | Ms - 3 digits, 0 decimals | xml. |
| | RAPDlog | 1 digit, 2 decimals | xml. |

For Pupil module, a typical continuous recording of the pupil size and parameters is shown below:



LogCon defined as  $-\log 10$  (contrast ratio), EG if the low brightness part of the stimulus is 2 nits, the high brightness part 255 nits, the LogCon would be  $-\log 10$  (2/255) =2, 1.

#### 5.1.2: Standard investigation

The supporting variables will be recorded by the Standard (ST) investigation for DR and AMD.

Table 3: The supporting variables with unit of the standard eye investigation

| Test | No of instances | Variable | Unit | Unit description |
|---|---|---|---|---|
| GAT | 1 | Pressure | mmHg | 2 digits, 1 decimal |
| iCare | 1 | Pressure | mmHg | 2 digits, 1 decimal |
| Acuity chart | 1 | Visual acuity | logMAR | 1 digit, 1 decimal |
| Contrast chart | 1 | Contrast acuity | Pelli-Robson score | 1 digit, 2 decimals |
| | 1 | Nasal step | | |
| | 1 | Temporal wedge | Present | |
| | 1 | Partial arcuate (sup) | | |
| | 1 | Partial arcuate (inf) | | Boolean |
| | 1 | Arcuate (sup) | | (true / false) |
| | 1 | Arcuate (inf) | | |
| | 1 | Altitudinal (inf) | | |
| | 1 | Altitudinal (sup) | | |
| | 1 | Paracentral | | |
| | | MD | dB | 2 digits, 2 decimals |
| Visual field | 54 | X coordinate | Degrees | 3 digits, 1 decimal |
| | | Y coordinate | Degrees | 3 digits, 1 decimal |
| | 1 | Threshold sensitivity | dB | 2 digits, 2 decimals |
| | 1 | Percentile degree | Score 1-5 | 1 digit |
| | 1 | Defuse defect | dB | 2 digits, 1 decimal |
| | 1 | Local defect | dB | 2 digits, 1 decimal |
| | 1 | sLV | dB | 2 digits, 1 decimal |
| | 1 | False positive | Percent (Reliability) | 2 digits |
| | 1 | False negative | Percent (Reliability) | 2 digits |
| | 1 | Mean Sensitivity | dB | 2 digits, 1 decimal |
| | 1 | Reliability factor | Percent (Reliability) | 2digits, 1 decimal |
| OCT RNFL | 1 | Average thickness | μm | 3 decimals |
| OCT GCL | 1 | Volume | mm^3 | 3 decimals |
| Pupil | 1 | Diameter change (max-min) | mm | 1 digit, 2 decimals |

The central variables related to DR and AMD will be "RAPD NDF", "Seen /unseen "," Time until the given point is recorded as seen", "the light in decibel when the point is seen", X- and Y-coordinates and "Pupil diameter in mm" and "OCT RNFL".

#### 5.2: Secondary variables

# 5.2.1: Quality-of- Life questionnaires<sup>30</sup>

The Quality-of-Life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded the same day as the first BCAM registration.

The QoL questionnaire EQ-5D-5L consists of 5 dimensions; "Mobility", "Self-care", "Usual activities", "Pain / Discomfort" and "Anxiety / Depression" <sup>30, 31, 32</sup>. Each of these five dimensions has 5 levels. Additionally, the patient scores the daily health situation on a 20 cm subdivided Visual Analogue Scale (VAS) with defined endpoints. The questionnaire is administrated by the investigators and will be given in patient's mother tongue language.

Under each heading or dimension, the patient is asked to describe the health situation today:

# MOBILITY I have no problems in walking about □ (1) I have slight problems in walking about □ (2)

BulbiCam; Validity study: V1\_OTH/DR; AMD-I/2022: Final Version 1.5\_22nd March 2022

| I have moderate problems in walking about I have severe problems in walking about I am unable to walk about | □ (3) □ (4) □ (5) |
|---|---|
| SELF-CARE I have no problems washing or dressing myself I have slight problems washing or dressing myself I have moderate problems washing or dressing myself I have severe problems washing or dressing myself I am unable to wash or dress myself | □ (1) □ (2) □ (3) □ (4) □ (5) |
| USUAL ACTIVITIES (e.g., work, study, housework, family or leisure a | ctivities) |
| I have no problems doing my usual activities | |
| I have slight problems doing my usual activities | $\square$ (2) |
| I have moderate problems doing my usual activities | $\Box$ (3) |
| I have severe problems doing my usual activities | $\Box$ (4) |
| I am unable to do my usual activities | $\Box$ (5) |
| PAIN / DISCOMFORT | |
| I have no pain or discomfort | $\Box$ (1) |
| I have slight pain or discomfort | |
| I have moderate pain or discomfort | |
| I have severe pain or discomfort | |
| I have extreme pain or discomfort | $\Box$ (5) |
| ANXIETY / DEPRESSION | |
| I am not anxious or depressed | |
| I am slightly anxious or depressed | |
| I am moderately anxious or depressed | |
| I am severely anxious or depressed | |
| I am extremely anxious or depressed | |

In addition, the patient will describe his /her daily health situation on a 100mm VAS (Figure 2)



Figure 2: EQ-Visual Analogue Scale

# 5.2.2: Common Terminology Criteria for Adverse Events version 4.0

The tolerability variables will be evaluated by using CTCAE version 4.0.<sup>33</sup> The CTCAE is divided in 26 System Organ Class (SOC) in accordance with the MedDRA hierarch. Within each SOC, adverse events (AE) are listed and accompanied by descriptions of severity or grade:

- Blood and lymphatic system disorders (11 Items)
- Cardiac disorders (36 Items)
- Congenital, familial, and genetic disorders (1 Items)
- Ear and labyrinth disorders (9 Items)
- Endocrine disorders (11 Items)
- Eye disorders (25 Items)
- Gastrointestinal disorders (117 Items)
- General disorders and administration site conditions (24 Items)
- Hepatobiliary disorder (16 Items)
- Immune system disorders (6 Items)
- Infections and infestations (76 Items)
- Injury, poisoning and procedural complications (77 Items)

- Investigations (38 Items)
- Metabolism and nutrition disorders (24 Items)
- Musculoskeletal and connective disorders (41 Items)
- Neoplasms benign, malignant, and unspecified incl. cysts and polyps (5 Items)
- Nervous system disorders (63 Items)
- Pregnancy, puerperium, and perinatal conditions (5 Items)
- Psychiatric disorders (20 Items)
- Renal and urinary disorders (20 Items)
- Reproductive system and breast disorders (51 Items)
- Respiratory, thoracic, and mediastinal disorders (59 Items)
- Skin and subcutaneous tissue disorders (34 Items)
- Social circumstances (2 Items)
- Surgical and medical procedures (1 Item)
- Vascular disorders (17 Items)

#### 5.2.2.1: Grading and classification of Items

Grade refers to the severity of the AE. The CTCAE displays Grade 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

Grade 0 = None

BulbiCam; Validity study:

Grade 1 = Mild: asymptomatic or mild symptoms; clinical or diagnostic

Observations only; intervention not indicated

Grade 2 = Moderate: minimal, local or non-invasive intervention indicated.

Limiting age-appropriate instrumental Activity of Daily Living (ADL)

Grade 3 = Severe or medically significant, but not immediately life-threatening:

Hospitalization or prolongation of hospitalization indicated disabling.

Limiting self-care ADL

Grade 4 = Life-threatening consequences; urgent intervention indicated

Grade 5 = Death related to AE.

Relationship to trial medication as: "Unrelated", "Possibly", "Probably" or "Definitely" Action taken as: "None"," Interruption", "Modified" or "Discontinued"

AE treatment as: "None", "Continue Medication", "Procedure" or

"Hospitalization"

Outcome at last visit as: "Resolved", "Ongoing" or "Fatal"

Definitions of relationship to study medication are as follows:

Unrelated: bears no relation to timing of medication, like symptoms or signs

expected in the disease process, does not recur on re-challenge.

Possibly: bears relation to timing of medication, like symptoms or signs expected

in the disease process, does not recur on re-challenge.

Probably: bears clear relation to timing of medication, distinct from symptoms or

signs expected in the disease process, does not recur on re-challenge.

Definitely: bears clear relation to timing of medication, distinct from symptoms or signs expected in the disease process, recurs on re-challenge.

#### 5.2.2.2: Outcome variables

The CTCAE results in two response variables. The main one is the sum of CTCAE score obtained by summarization of all the score obtained at a given visit. This is shown as Sum CTCAE. The second is the maximum) recorded score (Max CTCAE) given as the highest observed CTCAE score at a given visit. This is the most common way of reporting AE but has low statistical power to detect changes in toxicity during treatment. However, it is usable in classification of change in tolerability of treatment.

# 5.2.2.3: Serious Adverse Event (SAE)

An adverse event is any untoward symptom or sign befalling a patient in a clinical trial regardless of its relationship to the study medications. All adverse events must be described in detail and their severity and putative relationship to the study medication noted.

Adverse events may be considered seriously (SAE). The definition of this is as follows:

- Death
- Life threatening
- Leads to or prolongs hospitalization
- Results in persistent of significant disability
- Congenital anomaly

All adverse events will be recorded on relevant forms and their attribution to study medication will be evaluated. The severity of the reactions will be recorded along with a brief description of the event.

SAEs will be reported to sponsor and to the local sponsor representative via e-mail as soon as possible, but in any case, within 24 hours of the PI's knowledge of the event. It is the responsibility of the Principal Investigator to notify the Ethics Committee. It is the responsibility of the sponsor to report any Suspected Unexpected Serious Adverse Reactions (SUSAR) to the Regulatory Authority.

In case of SAE or SUSAR occurs, this will be handled in accordance with the hospital routines.

#### 5.3: Patient factors

BulbiCam; Validity study:

The patient factors recorded in the study will be age in days from birth to the screening visit calculated in the database and gender. The disease degree and previous and ongoing treatments of the disease will be recorded. Additionally, concomitant disease and treatments will be recorded.

Age and gender will be used to recruit controls to the included patients. Concomitant diseases and medication together with history of disease will be used to demonstrate the health condition of the participants at the time of inclusion in the study. Additionally, quality of life of the participants will be recorded at screening. This will also be a part of the health

evaluation but also gives the possibility of comparing the patients with the age- and gender matched controls.

# VI: Study procedure

# 6.1: Trial equipment and clinical procedure

In this study only Bulbicam (BCAM) version 1.7 will be used. Additionally, ST will be performed as the starting examination

The study will be performed according to European GCP regulation. All the participants have to perform BCAM registration twice per day in three consecutive days. Each registration will have duration of 15 minutes with one hour rest between the two observations. In case AE of grade 3 or 4 according to CTCAE occurs during the study, the participants will contact the responsible investigator. The BCAM registration will be stopped for at least 2 days or until the disappearance of the symptoms. The responsible investigator decides if the participant will continue or withdraw from the study.

#### 6.2: Inclusion visit and Screening phase

Both patients and the age- and gender matched controls must have a health situation in accordance with expectations related to the age and not suffering from other know serious disease. Participants, who fulfil the inclusion criteria; do not meet any of the exclusion criteria and willing to give informed consent to participate will be invited to participate and receive an appointment for starting the study (CRF III). No data from possible participants included in the screening phase but not fulfils the inclusion/exclusion criteria will be recorded in the database. During this initial inclusion visit, all demographic data and medical history will be recorded (CRF I & CRF II). Additionally, the QoL questionnaires EQ-5D-5L developed by EuroQol will be recorded initially as individual baseline values (CRF IV). The Common Terminology Criteria for AE (CTCAE) will be used for measuring the baseline AE situation (CRF V). The results from the initial measurements of the visual field and pupil obtained by ST will be recorded on CRF VI.

#### **6.3: Study procedure**

The clinical part of the study consists of two parts.

# 6.3.1: Part one (Repeatability)

This part will be performed the first day in the study; starting with the initial ST measurement and followed by two BCAM measurements (Fig 1). Each measurement includes the following six BCAM tests: Visual Field, Ptosis, Dynamic Acuity, Dynamic Contrast, Dark Adoption, and Pupil. Between the two measurements, a one-hour rest period will be included. ST includes Visual Field and Pupil. At the end of the last measurement a new CTCAE registration will be performed.

# 6.3.2: Part 2 (Stability)

This part will be performed during two following days and consists of two BCAM measurements each day (Fig 1). Each measurement includes the same six BCAM tests as described in part 1 with one-hour rest period between the two registrations. At the end of each day in this stability part a new CTCAE registration will be performed.

#### 6.4: End of the study

BulbiCam; Validity study:

As soon as possible after the last BCAM registration is done, the responsible investigator has to finalize the "End-of-Trial" CRF (CRF VI)

V1 OTH/DR; AMD-I/2022: Final Version 1.5 22<sup>nd</sup> March 2022

# 6.5: Stopping rule

If AE of grade 3 or 4 according to CTCAE occur, the participant will contact the responsible investigator. The BCAM registration will be stopped for at least 2 days or until disappearance of the symptoms. The responsible investigator decides if the participant will continue or withdraw from the study.

In case of life-threatening AE, SAE or SUSAR occurs, the BCAM registration has to stop until the disappearance of the symptoms. If possible, treatment of the symptoms will be given in accordance with the hospitals' routines. In case of life-threatening AE, SAE or SUSAR occurs at one of the sites, the other participating site will be informed at once by the study manager.

# 6.6: Report of serious adverse effect (SAE)

The patient will be advised to contact the investigator if she/he suffers from severe AE or any other annoying conditions.

In case of SAE or SUSAR, the investigator has to complete the SAE form and send it to the health authorities. All AE's will be recorded on relevant forms and their attribution to study intervention will be evaluated. The severity of the reactions will be recorded along with a brief description of the event.

SAEs and SUSAR will be reported to health authorities with copy to BulbiTech A/S and the project manager Prof. Stig Larsen by e-mail as soon as possible, but in any case, within 24 hours of the PI's knowledge of the event. It is the responsibility of the sponsor to report any SAE and SUSAR to the Regulatory Authority. In case of SAE or SUSAR occurs, this will be handled in accordance with the hospital routines.

Prof Stig Larsen
Meddoc AS,
Hvamstubben 14B 2013 Skjetten

Phone: +47 41 32 63 25 E-mail: sl@meddoc.no

#### 6.7: Study duration

BulbiCam; Validity study:

The study duration for each participant will be 3 days. The recruitment period is nine months. The time schedule of the study will be as follows:

| Inclusion of the first patient with control | 01-05-2022 |
|---------------------------------------------|------------|
| End of trial; last patient with control | 15-01-2023 |
| Closing database | 15-02-2023 |
| Finalized Clinical Study Report | 01-03-2023 |

# VII: Project management and Monitoring

#### 7.1: Project management

Prof Stig Larsen supported by Bård Dalhøi will administer the study. Vivy L Larsen (MSC) will oversee Data Management and clinical monitoring supported by the clinical staff at Meddoc. Hans E Fagertun (MSC) and Prof Larsen will oversee the statistical analysis. Prof Goran Petrovski will evaluate the ophthalmological part of the results.

#### 7.2: Publication of the results

The results will be published in an international medical journal. In principle, all the participating centers will be represented in the list of authors. The rules stated in the Vancouver recommendation will be followed.

#### 7.3: Quality assurance demands

The hospital sites will be monitored at regular intervals at site and electronically during the study. It is the duty of the investigator to provide open access to the monitor to all study related records at previously agreed times and locations.

In conducting the trial, the investigator accepts that the Sponsor, the regional Ethics Committee, the regulatory body, and monitor may, at any time, by appointment, conduct an audit of the study site.

In conducting the trial, the Sponsor accepts that the Ethics Committee or the regulatory body may, at any time, by appointment, conduct an audit of the study site, the laboratories conducting any clinical testing or the Good Manufacturing Practice (GMP) manufacturing facilities.

#### 7.4: Start-up and closing visit

The project manager and the clinical monitor will perform the start-up visit. The visit will consist of a site inspection, information, instruction and handing over the needed study materials as e-CRFs. A training program in use of the electronical data catching system InCRF will be given.

The project manager will perform the closing visit within one month after the last patient on the given site has finalized the study. All the trial material including CRFs will be removed from the site, but copies of the CRFs from the included patients will be stored at the site.

#### 7.5: Monitoring procedure

BulbiCam; Validity study:

Essential demographic data will be documented both within the patients' hospital record notes as source data and within the trial e-CRFs. This has to be available for inspection by the clinical trial monitor. Source data will also include the date of written consent. The times and dates of any other investigations must also be recorded.

It is the responsibility of the investigator to maintain accurate and up to date records of all clinical trial related activities, which should be legibly entered onto the e-CRFs provided. The e-CRFs should be made available to the monitor on request, and in the event of a formal investigator site audit.

On completion of the study, one copy of the e-CRFs will be retained at the hospital site for the duration stipulated by International Conference on Harmonization Good Clinical Practice (ICH/CGP), which currently is 5 years.

The eCRFs can be accessed online via web-based database InCRF. The contents of eCRFs should be approved by the investigators.

Monitoring at site will be performed at least three times at each participating hospital during the study. Monitoring report will be sent to the project manager latest one week after each site inspection.

#### 7.6: Curriculum vitae

The investigators have to submit an updated CV documenting their expertise in the relevant clinical field. The CV has to be signed and dated by the physician and a copy has to be attached to the protocol if required according to international rules. Another copy must be kept in the Trial Master File and a third copy in the Site File.

#### 7.7: Site file

BulbiCam; Validity study:

On behalf of the Sponsor, Meddoc AS will supply the investigators with a Site File. The Site File should contain all relevant documents for the study. The investigator is responsible for keeping the Site File updated and secure that all required documents are present in the Site File. The Site File will be inspected during the monitor visits.

# **VIII: Data Management**

#### 8.1. Case Record Forms (CRF)

In this study the electronical database and data catching system InCRF will be used. The identity of the participants in the database will be anonymized. The activation key is stored and only to be used by the clinically responsible ophthalmologist. Each study participants are given a study identification number which will be stored in the database. The data manager (DM) and the DM-staff at Meddoc will perform the secondary monitoring on the e-CRFs. Prior to study start, a data entry instruction document will be made. Source data consist of printouts from the laboratory examinations; baseline characteristics; clinical examination collected by the investigator and entered by site. In case of missing data or need of clarification, the responsible monitor will contact the site.

#### 8.2. Study Database

The validated data management system InCRF will be used for collecting the CRF data. The system selected is compliant with GCP guidelines and subject to 21 CFR (Code of federal regulations) FDA part 11 requirements. The final database will be stored in the Statistical Analysis system (SAS ver. 9.4 or later).

#### 8.3: Data handling

BulbiCam; Validity study:

A data entry person at site will enter the e-CRF data in InCRF and the DM will perform the initial data validation. In case of missing data, logical errors or interpretation problems, a query will be generated directly in InCRF. Investigator can review the query status via either InCRF function of "Study reports" /" Query report" or patient's e-Form dashboard. When all the needed participants have finalized the clinical part, and the investigator has electronically signed the e-CRFs, the DM will do the final verification checks and perform final database hard-lock when all errors are corrected.

Screening analysis for logical errors will be evenly performed on this database and errors will be corrected after new information is collected from the site. When all the detected errors are corrected, the main basic database will be locked. The database will be transformed to a labeled SAS database, which also will be locked up to prevent all possible changes or additions. In this copy, the responsible statistician can make derivations but no corrections of the data. If corrections are needed, the main basic study database has to be re-opened and corrected. The international procedure for such changes will be followed.

#### **IX:** Discontinuation

BulbiCam; Validity study:

A patient may discontinue the study at any time if, in the view of the investigator, it is in the participant's best interests. Alternatively, the participant has the right to discontinue her/his consent and exit the study without prejudice concerning her/his future treatment or care. If a participant does not show up to an agreed visit, the investigator should try to motivate her/him to continue. However, if the participant has decided not to continue, she/he should be asked to attend a control visit as described for the end of the study (CRF VI).

# 9.1: Discontinuation not related to the study question

A participant who discontinues the study for administrative reasons or reasons documented not related to the trial equipment classifies as "Drop out" and has to be replaced by a new participant. Such participants will not be included in the statistical analysis.

#### 9.2: Discontinuation related to the study question

Participants discontinue the study for the reasons are related to or might be related to the trial equipment will be classified as "Patient Withdrawal". These participants will not be replaced. They will be included in the Per-Protocol (PP) and the ITT analysis using the "Last-observation-carried-forward" (LOCF) procedure.

#### X: Ethical consideration

#### 10.1: Consideration of steering committee

The study will be conducted in compliance with the protocol and according to the Helsinki declaration with latest amendments and Good Clinical Practice (GCP).

Participants will only be included in this clinical trial after approval of the trial by the regional Ethical Committee (REK). The patients will receive oral and written information and have to give signed informed consent for participation.

All participants invited to participate in a clinical trial are entitled to make their decision based on the fullest amount of information available at that time. In order to make the choice, they will be given a written document expressed in a clear concise language of their native tongue to consider.

The document will tell potential participants about the nature of the measurements and the equipment. No interventions; only twice BCAM registration per day consecutively in three days. It will outline the numbers of participants in the trial, the steps of the protocol and type of measurements. This will give the participants a clear picture of the risks, inconveniences, and benefits that may accrue from the trial. The participants will be informed that she/he may decline the offer to join the trial or may withdraw at any time without prejudicing further medical care and is covered by the Sponsor's indemnity insurance in the event of mishap. Individuals must also know that their personal hospital records may be reviewed in confidence by the trial appointed research staff and that all personal information will be held on a confidential database. All information in the database will be anonymized and the activation key is stored by the clinically responsible ophthalmologist. Consent must always be given in writing after the participant has had time to reflect on the information and had an opportunity to ask further questions.

BCAM is new equipment, but certificated for clinical use [ISO 13485:2016] and sale in Norway (Appendix 15.2)

BCAM may increase the possibility for the investigator to give a safe diagnose at an early stage; give the final diagnose earlier and follow-up the patients more closely during treatment. However, before using such equipment in clinical practice the validity of the measurements must be documented.

*Summary:* No results from previous studies with this new equipment indicate any negative effect on the participants and AE has so far never been reported. All participants will be given oral and written information and have to give their written consent to participate in the study. To the best of our knowledge, this study fulfils the entire international requirement to an ethical controlled clinical trial.

#### 10.2: Approval of the project

BulbiCam; Validity study:

This study will be performed in Norway and the study protocol together and other requested information will be sent for approval by REK. Inclusion of patients will not be started before the approval is received.
The database and storage will be in Norway and must be approved by the Norwegian center for research data (NSD)

### 10.3: Informed consent

BulbiCam; Validity study:

Before the start of the trial, the investigator will explain the confidentiality of participation in this research project; the objectives of the trial; the specific requirements for the participating patients; the trial design and the consequences of participation. Additionally, the investigators have to obtain written informed consent from the participants before inclusion in the study.

### 10.4: Protection of personal data

The monitor may know the identity of the patients during verification of the source data. However, the monitor has unconditional professional secrecy.

All patient-related material leaving the department will be anonymous so that the patient only can be identified by date of birth, initials, and study number.

The investigator is responsible for keeping a list with the full names of the patients, their citizens' number, and corresponding study numbers according to the demands in GCP.

V1 OTH/DR; AMD-I/2022: Final Version 1.5 22<sup>nd</sup> March 2022

### XI: Statistical model

### 11.1: Handling of discontinuation

All patients fulfilling the inclusion and exclusion criteria, given informed consent to participate and started BCAM registration are classified as included in the study. In the ITT analysis, all these patients will be included and if necessary, the LOCF procedure will be used. The patients classified as Drop-out will be excluded from the statistical analysis.

### 11.2: Presentation of the result

Assumed continuously distributed variables will be expressed by mean values with 95% confidence intervals. <sup>34</sup> As an index of dispersion Standard Deviation (SD) will be used. The agreement index AI defined as AI=1 – [SD  $(X_1-X_2)$ /Mean  $(X_1-X_2)$ ] will be used for estimation of agreement in continuously variables and expressed by Blend & Altman plot. 35 Analysis of variance (ANOVA) with repeated measurements will be used in the analysis of stability. <sup>36</sup> In case of skewed distribution, the variable will be tried logarithmic transformed, and the analyses performed on the transformed data. The results will be retransformed for presentation. ANOVA will be used for comparison between patient groups and HC.<sup>37</sup> Categorized and discrete distributed variables will be expressed in contingency tables .<sup>38</sup>  $\kappa$ -analysis will be performed for estimation of agreement in these variables .<sup>39</sup> Additionally, important prevalence will be expressed in percentage with 95% confidence intervals constructed by using the theory of Simple Binomial Sequences.<sup>38</sup> Assumed continuously distributed variables will be expressed by mean values with 95% confidence intervals <sup>34</sup>. As an index of dispersion Standard Deviation (SD) will be used. In case of skewed distribution, the variable will be tried logarithmic transformed, and the analyses performed on the transformed data. The results will be retransformed for presentation.

Categorized and discrete distributed variables will be expressed in contingency tables.<sup>35</sup> Additionally, important prevalence will be expressed in percentage with 95% confidence intervals constructed by using the theory of Simple Binomial Sequences<sup>35</sup>.

### 11.3: Sample size

BulbiCam; Validity study:

With a significance level of 5%; a power of 90% and a Clinically Relevant Difference (CRD) of 1xSD between patient groups and HC, at least 16 HC and 16 patients in each diagnose have to be included.

### **XII: Operational matters**

### 12.1: Investigator's agreement

Before start, the investigators will confirm their agreements to participate in the trial by signing the Investigator's Agreement Form with the Sponsor.

#### 12.2: Instructions

The project manager, supported by the clinical monitor, will instruct the investigators at the start-up visit and during the study.

### 12.3: Amendments to the protocol

Changes in the protocol can be required by REK, investigators, project manager or Sponsor. Changes must be given in written amendments and numbered in the original protocol. It is forbidden to add new parameters consisting of measurements on the patients in the study unless they are covered as amendments in the protocol or taken due to the health and safety of the patient.

#### 12.4: Protocol deviations

Deviations from the protocol should be restricted as much as possible and will be fully recorded and justified. The project manager will be informed as soon as possible of all protocol deviations.

### **12.5:** Compliance monitoring

The project manager and the investigators will ensure that the site is suitable for the trial and that the participants are well informed of the particular trial. They shall check protocol compliance, handling of the test articles and recording of data during the critical stages of the trial. A report is prepared of each visit and kept in the trial master file (TMF).

### 12.6: Responsibilities

The investigators will acknowledge their responsibilities and their agreement to participate in the trial by dating and signing the agreement form. The project manager will verify that adequate arrangements have been made for the observations, measurements and recording of the data.

### 12.7: Confidentiality

BulbiCam; Validity study:

This clinical trial is a precondition for further studies in order to obtain permission to market the product worldwide. The Sponsor will therefore use the obtained data and results for the registration of the product. The main study database will be stored in the product database of the Sponsor.

The project manager and the investigators may demand and have the right to have the results published in an international medical journal. The draft of the manuscript has to be presented to the Sponsor for comments, discussion and final approval. The Sponsor cannot stop the

publication unless it is proved that publication of the results may damage the marketing of the product.

The project manager or the investigators cannot present the results in any meeting or congresses without approval by the Sponsor. The data obtained in this study has to be handled confidentially until the first registration of the product is performed.

### 12.8: Investigator and Sponsor withdrawals

BulbiCam; Validity study:

An investigator can finalize his or her participation in the study if BulbiTech A/S does not fulfill its duties according to the protocol or the Sponsor-investigator agreement. BulbiTech A/S has the right to terminate the study at any time. The investigators will be paid according to the agreements in the Sponsor-investigator agreement. A written explanation will be sent to all investigators and REK according to present rules.

### **XIII: References.**

- Council for International Organizations of Medical Sciences (CIOMS) guidelines. <a href="https://cioms.ch/shop/product/international-ethical-guidelines-for-health-related-research-involving-humans/">https://cioms.ch/shop/product/international-ethical-guidelines-for-health-related-research-involving-humans/</a>
- 2. Ting DS, Cheung GC, Wong TY. Diabetic retinopathy: global prevalence, major risk factors, screening practices and public health challenges: a review. Clin Exp Ophthalmol. 2016 May;44(4):260-77. doi: 10.1111/ceo.12696. Epub 2016 Feb 17. PMID: 26716602.
- 3. Teo ZL, Tham YC, Yan Yu MC, Chee ML, Rim TH, Cheung N, Bikbov MM, Wang YX, Tang Y, Lu Y, Hin Wong IY, Wei Ting DS, Wei Tan GS, Jonas JB, Sabanayagam C, Wong TY, Cheng CY. Global Prevalence of Diabetic Retinopathy and Projection of Burden through 2045: Systematic Review and Meta-analysis. Ophthalmology. 2021 Apr 30:S0161-6420(21)00321-3. doi: 10.1016/j.ophtha.2021.04.027. Epub ahead of print. PMID: 33940045.
- 4. Raman R, Rani PK, Reddi Rachepalle S, Gnanamoorthy P, Uthra S, Kumaramanickavel G, Sharma T. Prevalence of diabetic retinopathy in India: Sankara Nethralaya Diabetic Retinopathy Epidemiology and Molecular Genetics Study report 2. Ophthalmology. 2009 Feb;116(2):311-8. doi: 10.1016/j.ophtha.2008.09.010. Epub 2008 Dec 12. PMID: 19084275.
- 5. Pramanik S, Chowdhury S, Ganguly U, Banerjee A, Bhattacharya B, Mondal LK. Visual contrast sensitivity could be an early marker of diabetic retinopathy. Heliyon. 2020 Oct 26;6(10):e05336. doi: 10.1016/j.heliyon.2020.e05336. PMID: 33145449; PMCID: PMC7591734.
- 6. McAnany JJ, Park JC. Cone Photoreceptor Dysfunction in Early-Stage Diabetic Retinopathy: Association Between the Activation Phase of Cone Phototransduction and the Flicker Electroretinogram. Invest Ophthalmol Vis Sci. 2019 Jan 2;60(1):64-72. doi: 10.1167/iovs.18-25946. PMID: 30640972; PMCID: PMC6333111.
- 7. Park JC, Chau FY, Lim JI, McAnany JJ. Electrophysiological and pupillometric measures of inner retina function in nonproliferative diabetic retinopathy. Doc Ophthalmol. 2019 Oct;139(2):99-111. doi: 10.1007/s10633-019-09699-2. Epub 2019 Apr 23. PMID: 31016437; PMCID: PMC6742572.
- 8. Park JC, Chen YF, Blair NP, Chau FY, Lim JI, Leiderman YI, Shahidi M, McAnany JJ. Pupillary responses in non-proliferative diabetic retinopathy. Sci Rep. 2017 Mar 23;7:44987. doi: 10.1038/srep44987. PMID: 28332564; PMCID: PMC5362954.
- 9. Rukmini AV, Milea D, Gooley JJ. Chromatic Pupillometry Methods for Assessing Photoreceptor Health in Retinal and Optic Nerve Diseases. Front Neurol. 2019 Feb 12;10:76. doi: 10.3389/fneur.2019.00076. PMID: 30809186; PMCID: PMC6379484.
- 10. Jackson GR, Scott IU, Quillen DA, et al Inner retinal visual dysfunction is a sensitive marker of non-proliferative diabetic retinopathy British Journal of Ophthalmology 2012;96:699-703.
- 11. Bavinger JC, Dunbar GE, Stem MS, Blachley TS, Kwark L, Farsiu S, Jackson GR, Gardner TW. The Effects of Diabetic Retinopathy and Pan-Retinal Photocoagulation on Photoreceptor Cell Function as Assessed by Dark Adaptometry. Invest Ophthalmol Vis Sci. 2016 Jan 1;57(1):208-17. doi: 10.1167/iovs.15-17281. PMID: 26803796; PMCID: PMC4877135.
- 12. Klein R et al, Fifteen-year cumulative incidence of age-related macular degeneration: the Beaver Dam Eye Study, Ophthalmology 2007 Feb;114(2):253-62. doi: 10.1016/j.ophtha.2006.10.040.
- 13. Kahn HA et al, The Framingham Eye Study. I. Outline and major prevalence findings Am J Epidemiol 1977 Jul;106(1):17-32. doi: 10.1093/oxfordjournals.aje.a112428.
- 14. Bindewald A et al, Classification of abnormal fundus autofluorescence patterns in the junctional zone of geographic atrophy in patients with age related macular degeneration, Br J Ophthalmol 2005 Jul;89(7):874-8. doi: 10.1136/bjo.2004.057794.
- 15. Krishnan T et al, Prevalence of Early and Late Age-Related Macular Degeneration in India: The INDEYE Study, Invest Ophthalmol Vis Sci. 2010;51: 701–707) DOI:10.1167/iovs.09-4114.
- 16. Owsley C, Delayed Rod-Mediated Dark Adaptation Is a Functional Biomarker for Incident Early Age-Related Macular Degeneration, Ophthalmology, 2016 Feb;123(2):344-351. doi: 10.1016/j.ophtha.2015.09.041. Epub 2015 Oct 30.

- 17. Steinmetz RL, Haimovici R, Jubb C, et al. Symptomatic abnormalities of dark adaptation in patients with age-related Bruch's membrane change. Br J Ophthalmol. 1993; 77:549–54. [PubMed: 8218049]
- 18. Owsley C, Jackson GR, White MF, et al. Delays in rod-mediated dark adaptation in early age related maculopathy. Ophthalmology. 2001; 108:1196–202. [PubMed: 11425675]
- 19. Owsley C, McGwin G, Jackson G, et al. Cone- and rod-mediated dark adaptation impairment in age-related maculopathy. Ophthalmology. 2007; 114(9):1728–35. [PubMed: 17822978]
- 20. Dimitrov PN, Guymer RH, Zele AJ, et al. Measuring rod and cone dynamics in age-related maculopathy. Invest Ophthalmol Vis Sci. 2008; 49:55–65. [PubMed: 18172075]
- 21. Owsley C, Huisingh C, Clark ME, et al. Comparison of visual function in older eyes in the earliest stages of age-related macular degeneration to those in normal macular health. Curr Eye Res. 2015 E-pub ahead of print.
- 22. Hecht, S.; Shlar, S.; Pirenne, M.H. (1942). "Energy, Quanta, and Vision". Journal of General Physiology. 25 (6): 819–840. doi:10.1085/jgp.25.6.819. PMC 2142545. PMID 19873316.
- 23. Baylor, D.A.; Lamb, T.D.; Yau, K.W. (1979). "Responses of retinal rods to single photons". The Journal of Physiology. 288: 613–634. doi:10.1113/jphysiol.1979.sp012716 (inactive 2021-01-10). PMC 1281447. PMID 112243.
- 24. Stabell, U., and Stabell, B. (2003). Effects of light and dark adaptation of rods on specific-hue threshold. Vision Res. 43, 2905–2914. doi: 10.1016/j.visres.2003.07.003
- 25. Dimitrov PN, Robman LD, Varsamidis M, et al. Relationship between clinical macular changes and retinal function in age-related macular degeneration. Invest Ophthalmol Vis Sci. 2012;5213–5220.
- 26. Cocce KJ, Stinnett SS, Luhmann UFO, et al. Visual function metrics in early and intermediate dry age-related macular degeneration for use as clinical trial endpoints. Am J Ophthalmol. 2018;189:127–138.
- 27. Mollon JD. and Poldes PG. Post-Receptoral Adaptation, Department of Experimental Psychology, <u>Vision Research</u>, Volume 19, Issue 4, 1979, Pages 435-440
- 28. Reeves A, Distinguishing opponent and non-opponent detection pathways in early dark adaptation, Vision Research, 23 (1983), pp. 647-654
- 29. Reeves A, Grayhem R, Hwang AD, Rapid Adaptation of Night Vision, Department of Psychology, Northeastern University, Boston, MA, United States, Front. Psychol., 23 January 2018, https://doi.org/10.3389/fpsyg.2018.00008
- 30. EuroQol Group. EuroQol a new facility for the measurement of health-related quality of life. Health Policy 1990; 16:199 208
- 31. Herdman M, Gudex C, Lloyd A, Janssen MF, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D-5L. Quality of Life Research 2011 Dec; 20(10): 1727–36
- 32. Van Hout B, Janssen MF, Feng YS, Kohlmann T, Busschbach J, Golicki D, Lloyd A, Scalone L, Kind P, Pickard AS. Interim scoring for the EQ-5D-5L: mapping the EQ-5D-5L to EQ-5D-3L value sets. Value in Health 2012 Jul-Aug;15(5):708-15 doi:10.1016/j.jval.2012.02.008. Epub 2012 May 24
- 33. National Cancer Institute (NCI). Common Terminology Criteria for Adverse Events (CTCAE) version 4. June 2010: U.S. Department of Health and Human Service
- 34. Altman DG. Practical Statistics for Medical Research. Chapman & Hall, London 1999.
- 35. Bland JM, Altman DG (1986). "Statistical methods for assessing agreement between two methods of clinical measurement" Lancet. 327 (8476): 307–10
- 36. Girden ER. ANOVA; Repeated Measures. SAGE Publishing, Inc, California US 2001
- 37. Anderson TW. An Introduction to Multivariate Statistical Analysis. 3rd.Ed. John Wiley & Sons, New Jersey 2003.
- 38. Agresti A. Categorical Data Analysis. John Wiley & Sons, New Jersey 2002.
- 39. McHugh ML. Interrater reliability: the kappa statistic. Biochem Med (Zagreb). 2012 Oct; 22(3): 276–282.

### **XIV: Amendments**

### 14.1: Study identification

The Study identification has been changed from OTH /Dr; Amd; con - BCAM/ST - IM/1\_22 to V1 OTH/DR; AMD - I/2022

### 14.2: Study administration

The steering committee is specified page 1, point 0 to:

Project Manager: Professor Emeritus Stig Larsen; Norwegian University of Life

Sciences / Meddoc AS, Hvamstubben 14 2013 Skjetten

Project Coordinator: Bård Dalhøi. MSc Osteopathy

Chief Executive Officer (CEO) BulbiTech AS Trondheim

Responsible Ophthalmology: Professor Goran Petrovski Dr Med, MD, Ophthalmologist

Department of Ophthalmology, Oslo University Hospitals /

Ullevål Hospital, Oslo

PhD-fellow: Dr Bjørn Helland Hansen MD, Ophthalmologist

Department of Ophthalmology, Oslo University Hospitals /

Ullevål Hospital, Oslo

PhD supervisors: Prof Goran Petrovski and Prof Emeritus Stig Larsen

### 14.2: Specification of Standard examination

The specification of Standard examination is included in Chapter 1.7, 1.11, 2.3, and 5.2: The supporting variables will be recorded by the Standard (ST) investigation for DR and AMD.

| Test | No of instances | Variable | Unit | Unit description |
|---|---|---|---|---|
| GAT | 1 | Pressure | mmHg | 2 digits, 1 decimal |
| iCare | 1 | Pressure | mmHg | 2 digits, 1 decimal |
| Acuity chart | 1 | Visual acuity | logMAR | 1 digit, 1 decimal |
| Contrast chart | 1 | Contrast acuity | Pelli-Robson score | 1 digit, 2 decimals |
| | 1 | Nasal step | | |
| | 1 | Temporal wedge | | |
| | 1 | Partial arcuate (sup) | | |
| | 1 | Partial arcuate (inf) | | Boolean |
| | 1 | Arcuate (sup) | Present | (true / false) |
| | 1 | Arcuate (inf) | | (truc / faise) |
| | 1 | Altitudinal (inf) | | |
| | 1 | Altitudinal (sup) | | |
| Visual field | 1 | Paracentral | | |
| | | MD | dB | 2 digits, 2 decimals |
| | 54 | X coordinate | Degrees | 3 digits, 1 decimal |
| | | Y coordinate | Degrees | 3 digits, 1 decimal |
| | 1 | Threshold sensitivity | dB | 2 digits, 2 decimals |
| | 1 | Percentile degree | Score 1-5 | 1 digit |
| | 1 | Defuse defect | dB | 2 digits, 1 decimal |
| | 1 | Local defect | dB | 2 digits, 1 decimal |
| | 1 | sLV | dB | 2 digits, 1 decimal |

BulbiCam; Validity study: V1\_OTH/DR; AMD-I/2022: Final Version 1.5\_22nd March 2022

| | 1 | False positive | Percent (Reliability) | 2 digits |
|---|---|---|---|---|
| | 1 | False negative | Percent (Reliability) | 2 digits |
| | 1 | Mean Sensitivity | dB | 2 digits, 1 decimal |
| | 1 | Reliability factor | Percent (Reliability) | 2digits, 1 decimal |
| OCT RNFL | 1 | Average thickness | μm | 3 decimals |
| OCT GCL | 1 | Volume | mm^3 | 3 decimals |
| Pupil | 1 | Diameter change (max-min) | mm | 1 digit, 2 decimals |

The central variables related to DR and AMD will be "RAPD NDF", "Seen /unseen "," Time until the given point is recorded as seen", "the light in decibel when the point is seen", X- and Y-coordinates and "Pupil diameter in mm" and "OCT RNFL".

### 14.3: Study population

Chapter 3.2.1 is specified as: The study population 1 consists of patients diagnosed with DR of both gender; passed the age of 18 years; without any other eye disease; suffering from other know serious disease but have a health situation in accordance with expectations related to the age.

Chapter 3.2.2 is specified as: The study population 2 consists of patients diagnosed with AMD of both gender; passed the age of 18 years; without any other eye disease; suffering from other know serious disease but have a health situation in accordance with expectations related to the age.

Chapter 3.2.5 is specified as: The study population 3 consists of gender- and age-matched controls to patients in study population 1 or 2; passed the age of 18 years without any eye diseases; not suffering from other know serious disease and have a health situation in accordance with expectations related to the age.

Chapter 3.3 is specified as: No data from possible participants included in the screening phase but not fulfils the inclusion/exclusion criteria will be recorded in the database

Chapter 6.2 is specified with the following new introduction: Both patients and the age- and gender matched controls must have a health situation in accordance with expectations related to the age and not suffering from other know serious disease.

The following additional specification is done in *Chapter 6.2*: No data from possible participants included in the screening phase but not fulfils the inclusion/exclusion criteria will be recorded in the study database.

Chapter 5.2. The following information is added under 5.2.1: The Quality-of-Life (QoL) questionnaires EQ-5D-5L developed by EuroQol will be recorded once in the study and at the same day as the first BCAM registration. This will be performing as additional health verification and the possibility of comparing QoL of patients and controls.

### 14.4: Recruitment of patients

*Chapter 3.3* is rewritten and no given as follows:

The patients will be recruited from Oslo University hospital, Ullevål and Helgeland hospital. If necessary, private Ophthalmology clinics in Oslo will be asked for recruitment. All the investigations in the study will be performed by the same Ophthalmologist at the given hospital. The investigator informs the patients about the study, handing and collecting the written informed consent form. In case the patient fulfils the inclusion/exclusion criteria and willing to sign the consent form, the patient is included in the study. No data from possible participants included in the screening phase but not fulfils the inclusion/exclusion criteria will be recorded in the database. The included patient will be asked if he/she know any person with same gender and age; in good health condition without any eye disease which may participate as a control in the study. The potential controls will be contacted by the responsible investigator, obtain information about the study, and expected tasks. Controls willing to sign the consent form is included in the study. In case of lack in controls, requests among the hospital staff will be performed.

#### 14.5: Patient factor

The following paragraph are added to *chapter 5.5*: Age and gender will be used to recruit controls to the included patients. Concomitant diseases and medication together with history of disease will be used to demonstrate the health condition of the participants at the time of inclusion in the study. Additionally, quality of life of the participants will be recorded at screening. This will also be a part of the health evaluation but also gives the possibility of comparing the patients with the age- and gender matched controls.

### 14.6: Data Management

Additions to *Chapter 4.3*. All information in the database will be anonymized and the activation key is stored by the clinically responsible ophthalmologist.

Addition to *Chapter 8.1*. The identity of the participants in the database will be anonymized. The activation key is stored and only to be used by the clinically responsible ophthalmologist. Each study participants are given a study identification number which will be stored in the database

#### 14.7: Ethical consideration

BulbiCam; Validity study:

The previous statement under Chapter 10.1, page 34: "No results from previous studies with this new equipment indicate any negative effect on the participants and AE has so far never been reported" has been removed and replaced by "Despite that BulbiCam not previously has been used in any clinical study, it is nothing that may indicate that BulbiCam causes any adverse events.

The following specification is made in *Chapter 10.1*. All information in the database will be anonymized and the activation key is stored by the clinically responsible ophthalmologist

XV: Appendix

**15.1: Set of CRF's** 

BulbiCam; Validity study:

15.1.1: CRF I; Inclusion and exclusion

## Case Record Form I (A=DR)

(Inclusion and Exclusion criteria)

| Study | Study Id: V1_OTH /DR; AMD – I/2022; Participant Initials: | |
|---|---|---|
| Partic | Participant category. $DR$ patient $\square$ ; AMD patient $\square$ ; Healthy Control without any | |
| ophtha | almological or neurological disease | |
| <u>Inclus</u> | <u>ion criteria</u> | |
| A | Diagnosed with DR | $\square$ Yes $\square$ No |
| В | At least age of 18 years | $\square$ Yes $\square$ No |
| C | Without any other eye disease | □ Yes □ No |
| <u>Exclus</u> | sion criteria | |
| 1 | Other visual disturbances and blindness | □ Yes □ No |
| 2 | Posterior Chamber Artificial Ocular Lens (PCIOL) | $\square$ Yes $\square$ No |
| 3 | Physical or psychiatric disease disturbing the measuring procedure | e□ Yes□ No |
| 4 | Not able to perform full eye movements | $\square$ Yes $\square$ No |
| 5 | Visual acuity is less than 1 logMAR in any eye | $\square$ Yes $\square$ No |
| 6 | Visible part of the eye is abnormal. Haemorrhages/deformed pupil | $_{\mathrm{s}}\square$ Yes $\square$ No |
| 7 | Pupils not able to respond normally to dilation or contraction | $\square$ Yes $\square$ No |
| 8 | Participating another clinical trial with pharmaceuticals | $\square$ Yes $\square$ No |
| 9 | Not able to understand information | $\square$ Yes $\square$ No |
| 10 | With known alcoholic and drug dependency | $\square$ Yes $\square$ No |
| 11 | Not willing to give written consent to participate in the study | □ Yes □ No |
| Has the | e participant given written consent to participate? ☐ Yes ☐ No; Dat | te: 🗆 🗆 🗆 🗆 |
| Date: | Investigator (Sign) | |

# Case Record Form I (B=AMD) (Inclusion and Exclusion criteria)

| Stud | y Id: V1_OTH /DR; AMD – I/2022; Participant Initials: | |
|---|---|---|
| Part | icipant category. DR patient □; AMD patient □; Healthy C | ontrol without any |
| opht | halmological or neurological disease | |
| <u>Incl</u> | usion criteria | |
| A | Diagnosed with AMD | $\square$ Yes $\square$ No |
| В | At least age of 18 years | $\square$ Yes $\square$ No |
| C | Without any other eye disease | □ Yes □ No |
| <u>Excl</u> | usion criteria | |
| 1 | Other visual disturbances and blindness | ☐ Yes ☐ No |
| 2 | Posterior Chamber Artificial Ocular Lens (PCIOL) | $\square$ Yes $\square$ No |
| 3 | Physical or psychiatric disease disturbing the measuring proced | ure 🗆 Yes 🗆 No |
| 4 | Not able to perform full eye movements | $\square$ Yes $\square$ No |
| 5 | Visual acuity is less than 1 logMAR in any eye | $\square$ Yes $\square$ No |
| 6 | Visible part of the eye is abnormal. Haemorrhages/deformed pu | pils□ Yes □ No |
| 7 | Pupils not able to respond normally to dilation or contraction | $\square$ Yes $\square$ No |
| 8 | Participating another clinical trial with pharmaceuticals | $\square$ Yes $\square$ No |
| 9 | Not able to understand information | $\square$ Yes $\square$ No |
| 10 | With known alcoholic and drug dependency | $\square$ Yes $\square$ No |
| 11 | Not willing to give written consent to participate in the study | □ Yes □ No |
| Has | the participant given written consent to participate? $\square$ Yes $\square$ | ] No; Date: □□ □□ □□ |
| | | , |
| | 1 (0: ) | |
| Date | Investigator (Sign) | |

BulbiCam; Validity study:

## 15.1.2: CRF II; Demographic factors

# Case Record Form II (Demographic factors)

| Study Id: V1_OTH/DR; AMD-I/2022 [Transferred from the system] |
|---|
| Country: ☐ (Norway=1; India=2 etc); Site: ☐ (First site =1 Second=2 etc); Disease ☐ (None =0; |
| Glaucoma=1; Cataract=2; DR =3 etc); Disease degree ☐ (None=0; Mild =1; Moderate =2; Severe=3); |
| Running number: $\square\square$ [Created from the system within the group defined by information above] |
| Participant Id-number: \[ \bigcap \Bigcap \Big |
| Patient initials; Date of inclusion: $\Box\Box\Box\Box\Box\Box\Box$ |
| Demographic factors |
| Date of birth: $\square$ $\square$ $\square$ $\square$ Age: $\square$ (years), Gender: $\square$ (Male=M; Female=F) |
| Comment: |
| Comment. |
| Investigator (Sign) Date: |

BulbiCam; Validity study:

## 15.1.3: CRF III; Medical history

## Case Record Form III (A=DR)

(Medical history)

| Study Id: V1_OTH/DR; AMD-I/2022[Transferred from the system] |
|---|
| Participant Id-number: \[ \Bigcup \Big |
| 1 . 1 7: |
| <u>Actual disease</u> |
| Specification: DR; Date first time diagnosed: □□ □□ □□ |
| Degree (classification) of disease: ☐ [specification for each study] |
| Ongoing treatment |
| Date of start: |
| Ongoing concomitant disease |
| □Gastrointestinal, □General disorders, □Hepatobiliary, □Immune system disorder □Infections, □Injury and procedural, □Investigations, □Metabolism and nutrition, □Musculoskeletal, □Neoplasm, □Neurology, □Ophthalmology, □Pregnancy and perinatal, □Psychiatric, □Renal and urinary, □Reproductive, □Respiratory, □Rheumatic, □Skin, □Social circumstances, □Surgical and Medical, □Vascular |
| Ongoing concomitant diagnoses |
| Ongoing concomitant treatment |
| Date of start: □□ □□□□□ Date of start: □□ □□□□□ |
| Date of start: |
| Date of start. |
| Date: □□ □□ □□ |

## Case Record Form III (B=AMD)

(Medical history)

| Study Id: V1_OTH /DR; AMD – I/2022 [Transferred from the system] |
|---|
| Participant Id-number: \[ \Bigcup \Big |
| Actual disease |
| Specification: AMD; Date first time diagnosed: $\Box\Box\Box\Box\Box\Box$ |
| Degree (classification) of disease: ☐ [specification for each study] |
| Ongoing treatment |
| Date of start: □□□□□□ Date of start: □□□□□□ Date of start: □□□□□□ Date of start: □□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□□ |
| Ongoing concomitant disease |
| □ Gastrointestinal, □ General disorders, □ Hepatobiliary, □ Immune system disorder □ Infections, □ Injury and procedural, □ Investigations, □ Metabolism and nutrition, □ Musculoskeletal, □ Neoplasm, □ Neurology, □ Ophthalmology, □ Pregnancy and perinatal, □ Psychiatric, □ Renal and urinary, □ Reproductive, □ Respiratory, □ Rheumatic, □ Skin, □ Social circumstances, □ Surgical and Medical, □ Vascular Ongoing concomitant diagnoses |
| Ongoing concomitant treatment |
| Date: \( \sum |

BulbiCam; Validity study:

## 15.1.4: CRF IV; Quality of life

BulbiCam; Validity study:

## Case Record Form IV (Quality of Life)

| Study Id: V1_OTH /DR; AMD – IM/1_22 [Transferred from the sys | stem] |
|---|---|
| Participant Id-number: \[ \Bigcup \Bigcup \Bigcup \Bigcup \Bigcup \Bigcup \Interpooling Transferred from CRF I] | |
| EQ-5D-5L | |
| BEVEGELSE Jeg har ingen problemer med å gå rundt Jeg har noen problemer med å gå rundt Jeg har moderate problemer med å gå rundt Jeg har store problemer med å gå rundt Jeg klarer ikke å gå rundt | □ (1)<br>□ (2)<br>□ (3)<br>□ (4)<br>□ (5) |
| SELVPLEIE Jeg har ingen problemer med å vaske eller kle på meg Jeg har noen problemer med å vaske eller kle på meg Jeg har moderate problemer med å vaske eller kle på meg Jeg har store problemer med å vaske eller kle på meg Jeg klarer ikke å vaske eller kle på meg | □ (1)<br>□ (2)<br>□ (3)<br>□ (4)<br>□ (5) |
| VANLIGE AKTIVITETER (f.eks. arbeid, studier, husarbeid og familie Jeg har ingen problemer med å gjøre de vanlige aktivitetene mine Jeg har noen problemer med å gjøre de vanlige aktivitetene mine Jeg har moderate problemer med å gjøre de vanlige aktivitetene mine Jeg har store problemer med å gjøre de vanlige aktivitetene mine Jeg klarer ikke å gjøre de vanlige aktivitetene mine | - eller fritidsaktiviteter) (1) (2) (3) (4) (5) |
| SMERTER / UBEHAG Jeg har ingen smerter eller ubehag Jeg har noen smerter eller ubehag Jeg har moderate smerter eller ubehag Jeg har store smerter eller ubehag Jeg har ekstrem smerte eller ubehag | ☐ (1)<br>☐ (2)<br>☐ (3)<br>☐ (4)<br>☐ (5) |
| ANGST / DEPRESSJON Jeg er ikke engstelig eller deprimert Jeg er noe engstelig eller deprimert Jeg er engstelig eller deprimert Jeg er veldig engstelig eller deprimert Jeg er ekstremt engstelig eller deprimert | □ (1) □ (2) □ (3) □ (4) □ (5) |

## **EQ-Visual Analogue Scale (VAS)**

Pasienten skal beskrive sin daglige helsesituasjon på en 100mm VAS ved å avsette en horisontal strek på skalaen nedenfor hvorav «0» angir «Den verste helsen du kan forestille deg» og «100» angir «Den beste helsen du kan forestille deg»

Angi resultatet i mm fra bunnen og opp til merket på skalaen nedenfor: □□□mm

## The best health you can imagine

The worst health you can imagine

## Case Record Form V

(Adverse Event)

| Study Id: V1_OTH /DR; AMD – I/2022 | [Transferred from the system] |
|------------------------------------|-------------------------------|
|------------------------------------|-------------------------------|

| Participant Id-number: | $\square \square$ [Trans | sferred from | CRF I |
|------------------------|--------------------------|--------------|-------|
|------------------------|--------------------------|--------------|-------|

| Adverse<br>Event (specify | <b>Severity</b> (1 - 5) | SAE<br>(N/Y) | Relationship to medical device | Action taken | AE<br>treatment | Date<br>Started | Date<br>Stopped | Outcome (1-3) |
|---|---|---|---|---|---|---|---|---|
| ) | | | (1-4) | (1-4) | (1-4) | (ddmmyy) | (ddmmyy) | |

| Classifications | | | | | |
|---|---|---|---|---|---|
| Severity of AE | SAE | Relationship to IP | Action Taken | AE Treatment | Outcome |
| 1 = Mild<br>2 = Moderate<br>3 = Severe<br>4 = Life<br>threatening<br>5 = Death | N = No<br>Y = Yes | 1 = Unrelated 2 = Possibly 3 = Probably 4 = Definitely | 1 = None 2 = Interruption 3 = Modified 4 = Discontinued | 1 = None<br>2 = Continue<br>Medication<br>3 = Procedure<br>4 = Hospitalization | 1 = Resolved<br>2 = Ongoing<br>3 = Fatal |

## 15.1.6: CRF VI; Adverse Events

## **Case Record Form VI**

(Initial registration by ST)

| Study Id: V1_OTH /DR; AMD–I/2022 [Transferred from the system] | |
|---|---|
| Participant Id-number: \[ \Bigcup \Big | |
| The Standard method | |
| GAT-pressure: iCare-pressure: Acuity chart: Contrast chart: Visible Field Point seen: Nasal step: Temporal wedge: Partial arcuate (sup): Partial arcuate (inf): Arcuate (sup): Arcuate (inf): Altitudinal (inf): Altitudinal (sup): Paracentral: | □□,□ mmHg □,□ mmHg □,□ mmHg □,□ mmHg □Yes □No □Yes □No |
| MD: X-coordinate Y-coordinate Threshold sensitivity Percentile degree Defuse defect Local defect sLV False positive False negative Mean Sensitivity | □□□,□ dB □□,□□ degree □□,□ dB □ Score (1 – 5) □□,□dB □□,□dB □□,□dB □□,□dB □□,□dB □□,□dB |
| OCT RNFL:<br>OCT GCL:<br>Pupil diameter size: | $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ |
| Date: | Investigator's signature: |

## 15.1.7: CRF VII; End of Trial

BulbiCam; Validity study:

## Case Record Form VII (End of Trial)

| • | Id: V1_OTH /DR; AMD–I/2022 [Transferred from the system] ipant Id-number: \[ \Bigcap \ |
|---|---|
| Please | e state the trial end reason: |
| | Completion of trial |
| | Withdrawal: patient withdrew consent. |
| | Date withdrawal (dd-mm-yyyy): |
| | Reason withdrawal: |
| | □ Adverse experience – please specify: |
| | ☐ Inter-current illness (must be reported as an AE) |
| | ☐ Protocol Violation- please specify: |
| | Drop-out: patient request. |
| | Date drop-out (dd-mm-yyyy): |
| | Patient lost to follow up. |
| | Date last contact (dd-mm-yyyy): |
| | <b>Death</b> – must be reported as a SAE. |
| | Date of death (dd-mm-yyyy): |
| | Other, please specify: |
| | Date of discontinuation (dd-mm-yyyy): |
| I hereb<br>comple<br>dates s | by certify that the entries on all pages of this Case Report Form accurately and etely represent the results of the examinations, tests, and evaluations performed on the specified. |
| Date: | Investigator's signature: |

### 15.2: Bulbicam Certificate

15.2.1: ISO-Certificate



### 15.2.2: Certificate of free Sales



To Whom it May Concern

NO-20/11005

Date: 08.02.2021

#### Certificate of Free Sales

The Norwegian Medicines Agency as Competent Authority for medical devices hereby certifies that the products listed below are manufactured by:

Bulbitech AS Krambugata 2 7011 Trondheim Norway

We have been notified that the following medical devices are sold as CE-marked products:

| Cat. Number | Product Name |
|-------------|-------------------------------------------------------------|
| 65177 | BulbiCAM - Vision physiology / eye movement analysis system |

The precondition for medical devices to be CE-marked in compliance with directive 90/385/EEC, directive 93/42/EEC or directive 98/79 EC is to meet the essential requirements for safety. A CE-marked medical device may therefore be placed on the market in Norway without any approval from the Medicines Agency and may be exported without any restrictions.

This certificate is valid until 08. February 2023

Raymond Ludvigsen Segior Adviser

Consultant

Norwegian Medicines Agency (NoMA)
Festbeks 240 Skøyen 0213 Cbb, Norwey
Vist address, Gensensinger 26, 1868 Oslo, Norway
post@nome.no or medevi-ru@nume.no
noma.no

Letters should be adressed to the Norwegian Middletes. Agency Places state our reference. Tit. 447,22,83,77,00 (2ANL: NO.71,764,65,65). SWFT, DNBANCKK.

## 15.3: CV; Primary investigator & Steering Committee

### 15.3.1: Bård Dalhøi CEO BulbiTech AS

### **Curriculum vitae**

### \* PERSONAL INFORMATION

| *Family name, First name: | Dalhøi, Bård | | |
|---------------------------|--------------|-------|------|
| *Date of birth: | 18.06.64 | *Sex: | Male |
| *Nationality: | Norwegian | | |

### \* HIGHER EDUCATION/OTHER TRAINING

| | Subjects/degree/ | Name of institution, country |
|---|---|---|
| 1987-1989 | Physical Therapy | REHA-Zentrum Berlin |
| 1990-1995 | Diploma degree in Osteopathy | Norwegian Academy of Osteopathy |
| 2007-2008 | Medical PhD studies in<br>Medical Research<br>Methodologies | NMBU – Norwegian University of Life Sciences |
| 2008 | Medical PhD studies in<br>Experimental design in<br>clinical studies | Faculty of Life Sciences, University of Copenhagen |

<sup>\*</sup> POSITIONS (academic, business, industry, public sector, national or international organisations)

### **Current Position**

| Job title/name of employer/country | |
|---|---|
| 2021- | Chief Executive Officer, Bulbitech AS |
| 2015 - | Chief Scientific Officer, BulbiTech AS, Norway |
| 2013-2015 | Chief Executive Officer, Bulbitech AS, former Heads AS, Norway from 2013-2019 |

### Previous positions held (list)

| Job title/nar | ne of employer/country |
|---|---|
| 1995-2013 | Private Practice and co-founder, Osteopatiklinikken Midt-Norge AS, Norway |

BulbiCam; Validity study: V1\_OTH/DR; AMD-I/2022: Final Version 1.5\_22nd March 2022

| 2010-2012 | Senior lecturer, Program Osteopathy, Høyskolen Kristiania, Norway |
|---|---|
| 1997-2010 | Co-founder of Academy of Osteopathy, board member and lecturer in Program for Osteopathy Nordic Academic of Osteopathy, Norway |
| 1990-1997 | Private Practice, Fjordgata Fysioterapi & Osteopati, Norway |
| 1993-1995 | Clinical lecture, Physical therapy, University NTNU, Norway |
| 1989-1990 | Clinical practice, Physical Therapy department, St. Olav Hospital, Norway |

### **PROJECT MANAGEMENT EXPERIENCE**

BulbiCam; Validity study:

| Project/topic/role in project/funding from | |
|---|---|
| 2021- | Project leader BulbiEYE. Project was approved in Norwegian Research Council June 2021. Budget 20 mNOK. |
| 2015-2020 | Development of the first version of hardware (BulbiCAM) and software (BulbiHUB) – patent BulbiCAM, public funding application and project leader: 3 major projects supported by Innovation Norway 2015-2018 LASFIN, 2016-2017 HASFIN, 2019-2020 Project BulbiCAM and SkatteFunn LASFIN and HASFIN |

### **EXPERIENCE FROM RELEVANT RESEARCH & INNOVATION ACTIVITIES** (if applicable)

| Project/type of R&I activity and R&I content /role and tasks/funding from | |
|---|---|
| 2018- 2019 | Publications: |
| | Randomized two dimensional between patient response surface |
| | pathway design with two interventional and one response variable in estimating minimum efficacy dose, International Journal of Clinical |
| | Trials |
| | 2. Osteopathic manual Therapy (OMT) in treatment of gastroesophageal reflux |
| | disease (GERD), Larsen S et al. Int J Clin Trials. 2019 Aug;6(3):75-83, Clinical |
| | Practice. |
| 2017 | Chennai, India Sankara Nethralaya Glaucoma Meet (SANGAM) September 2017 |
| | Binocular pupillometry: Quantification of pupillary responses using eye tracking technology |
| 2017 | Hyderabad, India World Congress of Optometry (WCO) 2017Clinical applicability of an |
| | eye tracker based pupillometry system |
| 2017 | VISION conference June 2017 |
| | An approach to quantify the pupil response using an eye tracker-based pupilometer |

### **EXPERIENCE FROM NATIONAL/INTERNATIONAL COLLABORATION/NETWORKING** (if applicable)

Activity or project / tasks and responsibilities / context/programme/framework of the collaboration and names of key partners (companies, institutions)

| 2021-2023 | Project leader of BulbiEYE, granted from Norwegian Research Council. Project partners: Collaborating partners; Oslo University Hospital (Ullevål Eye Dept and Rikshospitalet Nero Dept), Helgelandssykehuset Eye Dept., Meddoc AS |
|---|---|
| 2021- | Clinical validation of Eye Movement based Acuity, Contrast and Dark Adaptation test. Pupil RAPD test, Vergence test, Nystagmus test. |
| 2020 | Study measuring the reliability, and stability of Video Oculography Device in BulbiCAM in |
| | Eye Movement Perimetry and Pupillometry. Coordinator and study leader of the overall study's progress in collaboration with the Medical Research Foundation at Sankara Nethralaya Eye Hospital (India) and Prof. Emeritus Stig Larsen at Meddoc AS (Norway). |
| 2019-2020 | Clinical validation of eye tracking, pupillometry and nystagmography (Pupil, Visual Field, Saccades, Ptosis, Worth 4 dot, Amsler test); coordinator and study leader of the overall study's progress; collaboration with the Medical Research Foundation/Sankara Nethralaya Eye Hospital (India), Ass Prof Johan Pel, Department of Neuroscience, Erasmus MC, The Netherlands, and Prof. Stig Larsen, Norwegian University of Life Science. |
| 2015-2018 | Project leader, LASFIN project partners: Neuroscience department at Erasmus MC, NL, EyeSeeTech Gmbh, Munich, Germany, Lameris Ootech BV, NL, Medical Research Foundation, Sankara Nethralaya Eye Hospital, Chennai, India |

### OTHER MERITS RELEVANT TO THE PROJECT

BulbiCam; Validity study:

- Project manager of BulbiEYE project, which is a 2 mill. Euro industrial and clinical projects financial supported by the Norwegian Research Council
- Project manager of 3 Innovation Norway financial supported projects
- Publications, technical reports, peer-review assignments, etc.
- Presentations at workshops or conferences (national/international level)
- Positions in professional associations/networks

Bård is the CEO and CSO at BulbiTech AS with a working experience within the biotechnology industry and has experience in clinical research, including the development and participation in studies concerning the osteopathic clinical research and clinical research in medical technology development. Bård is skilled in clinical research, pain management, healthcare, rehabilitation, and sports medicine. His work has brought him in contact with several research institutions, enabling him to increase its network for national and international collaborations. His experience within the medical field and clinical care goes back to 1989, when Bård started his professional practice as a Physical Therapist in both public and private hospitals and clinics, and from 1995 as an Osteopath at private healthcare institutions. Co-founder and chairman Norwegian Association of Osteopathy founded 09.06.1997, which was public registered 15.07.1997. Cofounders and board member of the Norwegian Academy of Osteopath. Today the education is approved as a health care education with a BSc degree, and the profession is to get their official authorisation in Norway 2021. Since 2013, Bård was the co-founder of Bulbitech AS (former Heads AS) and served as a CEO in Heads from 2013 until 2015. Re-engaged as a CEO in Bulbitech in 2021 and holds both the position as a CEO and CSO (Chief Science Officer).

## 15.3.2: Professor Goran Petrovski; Ophthalmology

**Role in the project** Project manager ⊠ Project partner □

### **Personal information**

| First name, Surname: | Goran Petrovski | | |
|---|---|---|---|
| Date of birth: | 13.02.1975 | Sex: | M |
| Nationality: | Hungarian | | |
| Researcher unique identifier(s) (ORCID, ResearcherID, etc.): | 0000-0003-2905-9252 | | |
| URL for personal website: | https://www.med.uio.no/klinmed/personer/vit/goranpe/index.html | | |

### **Education**

| Year | Faculty/department - University/institution - Country |
|---|---|
| 2007 | Ph.D. |
| (dissertation defended) | University of Debrecen, Medical and Health Science Center (UDMHSC), Dept. of Biochemistry and Molecular Biology , Hungary |
| 2003 | Medical Doctor |
| | UDMHSC, Hungary |

### **Positions - current and previous**

| Year | Job title – Employer - Country |
|---|---|
| 2016- | Professor and Head of the Center of Eye Research, Department of Ophthalmology,<br>Oslo University Hospital and UiO, Oslo, Norway |
| 2013-2016 | Associate Professor of Ophthalmology and Head, Stem Cells and Eye Research Laboratory, Department of Ophthalmology, University of Szeged, Hungary |

## Project management experience

BulbiCam; Validity study:

| Year | Project owner - Project - Role - Funder |
|---|---|
| 2020-2023 | Principal investigator/project leader – "Optimization of stem cell-laden smart biomaterials for 3D bioprinting of human cornea" – Norway-India collaborative project – Funder: Norwegian Research Council |
| 2021-2024 | Principal investigator/project leader – "Development of standardized culture, transplantation and banking of RPE cells for treatment of age-related macular degeneration (AMD)" – Norway-Czechia collaborative project – Funder: EEA Norway grants |

### 15.3.3: Professor Stig Larsen

## Curriculum vitae (CV) with track record

| Role in the project | Manager $\square$ | Partner | $\boxtimes$ |
|---------------------|-------------------|---------|-------------|

### **Personal information**

| First name, Surname: | Stig Larsen | | |
|---|---|---|---|
| Date of birth: | 26.March 1947 | Sex: | Male |
| Nationality: | Norwegian | | |
| Researcher unique identifier(s) (ORCID, Researcher ID, etc.): | 0000-0001-9591-9324 | | |
| URL for personal website: | | | |

### **Education**

| Year | Faculty/department - University/institution - Country |
|---|---|
| 1982 | PhD: Dept. of Gastroenterology/Ullevål Hospital- Oslo University -Norway |
| 1975 | Cand. Real: Dept. of Mathematics/Master- Oslo University -Norway |

### **Positions - current and previous**

| Year | Job title – Employer - Country |
|---|---|
| 2017- | - Prof Emeritus- Norwegian University of Life Sciences (NMBU)- Norway - Research Director- Meddoc-Norway |
| 2000-2017<br>1990-2000<br>1990-2000 | -Professor I; Controlled clinical Research Methodology- NMBU- Norway -Professor II: Norwegian School of Veterinary Medicine-Norway -Research Director: Medstat/Parexel- Europe |

### **Project management experience**

(Academic sector/research institutes/industrial sector/public sector/other. Please list the most relevant.)

| Year | Project owner - Project - Role - Funder |
|---|---|
| 2018-2020 | Tine SA- The effect of optimized daily intake of Jarlsberg cheese on s-Osteocalcin and Vitamin K2- Project manager. [Publication 10; reference list]. |
| 2020- 2022 | Tine SA- Comparison of Jarlsberg® cheese and cheese without content of vitamin K2 on s-Osteocalcin- Project manager. [NFR-IPN project; Additionally, 3 manuscripts under preparation for international publication] |

BulbiCam; Validity study: V1\_OTH/DR; AMD-I/2022: Final Version 1.5\_22nd March 2022

### **Supervision of students**

| Master's students | Ph.D.<br>students | University/institution - Country |
|---|---|---|
| 1 | 16 | NMBU/Faculty of Veterinary Medicine -Norway |
| 0 | 12 | Oslo University/ Faculty of Medicine-Gastroenterology-Norway |
| 1 | 1 | Bergen University/ Faculty of Medicine- Rheumatology-Norway |
| 0 | 2 | Oslo University/ Faculty of Medicine- Radiology-Norway |
| 2 | 3 | Norwegian School of Sport Science-Norway |
| 5 | 0 | Norwegian School of Osteopathy |

### Other relevant professional experiences

| Year | Description - Role |
|---|---|
| 1992 - 2000 | Research Manager; Development of PTW-design: An Adaptive design approach. |
| | [Publication 1-3; Additionally 4 international papers are published + 1 PhD] |
| 2000 - 2020 | Research Manager; Development of Response Surface Pathway (RSP) design. |
| | [Publication 4-6; Additionally, 11 paper are internationally published + 2 PhD] |
| 2003 | Research Manager; The effect of an Ergonomic Intervention on Musculoskeletal, |
| | Psychosocial and Visual Strain of VDT Entry Work: Organization and Methodology of |
| | International Study. [Publication 7; Additionally, 4 papers are internationally |
| 2010 – 2020 | published] |
| | Research Manager; Clinical documentation of a new immune modulating |
| | chemotherapeutic drug (BP-C1) in treatment of breast cancer and gastric cancer. |
| 2018 - 2022 | [Publication 5,8 and 9; Additionally 8 papers are internationally published] |
| | Project Manager; The effect of daily Jarlsberg cheese intake on the Osteocalcin level |
| | and vitamin K2 status to healthy premenopausal women. [Publication 10; Additionally |
| | 3 more manuscripts ready for evaluation in international journals ] |

### **Track record**

## A: 342 scientific publications in international peer-reviewed journals; 10 related publications given

- Reiertsen O, Larsen S, Størkson R, Trondsen E, Løvig T, Andersen OK, Lund H & Mowinckel P. Safety of enoxaparin and dextran 70 in the prevention of venous thromboembolism in digestive surgery. A Play-the-Winner designed study. Scand.J.Gastroenterol. 1993; 28:1015-1020.
- 2) Larsen S, Reiertsen O, Mowinckel P, Lund H & Osnes M. Play The Winner: a step-by-step process design to compare and control the efficacy and safety of treatments. Pharm. Med. 1994; 8: 11-23.

BulbiCam; Validity study: V1\_OTH/DR; AMD-I/2022: Final Version 1.5\_22<sup>nd</sup> March 2022

- 3) Bjerkeset O, Larsen S & Reiertsen O. Evaluation of enoxaparin given before and after operation to prevent venous thrombo-embolism during digestive surgery: Play-the-Winner designed study. World J Surg 1997; 21: 584-589.
- 4) Dewi S; Aune T, Buanæs JAAa; Smith A; Lasen S. The development of response surface pathway design to reduce animal number in toxicity studies. BMC Pharmacology and Toxicology, 2014; 15: 18-28
- 5) Dewi S; Kristiansen V; Lindkær-Jensen S & Larsen S. Between Patient, n-level Response Surface Pathway Design in dose-finding studies. Open Access Journal of Clinical Trials, 2014; 6: 1-12.
- 6) Larsen S, Holand T, Bjørnæs KE, Glomsrød E, Kaufmann J, Garberg TH, Elvbakken G, Dalhøi B, Reiertsen O & Dewi S. Randomized two-dimensional between-patient Response Surface Pathway design with two interventional- and one response variable in estimating Minimum Efficacy dose. Int J Clin Trials. 2019 Aug; 6(3):75-83.
- 7) Dainoff M, Aarås A, Horgen G, Konarska M, Larsen S, Thoresen M, Cohen BGF. The Effect of an Ergomic Intervention on Musculoskeletal, Psychosocial and Visual Strain of VDT Data Entry Work: Organization and methodology of the international study. JOSE 2005; 11 (1): 9-23.
- 8) Larsen S; Butthongkomvong K; Manikhas A; Trishkina E; Poddubuskaya E; Matrosova M; Srimuninnimit V; Lindkær-Jensen S. BP-C1 in the treatment of patients with stage IV breast cancer: a randomized, double-blind, placebo-controlled multicentre study and an additional open-label treatment phase. Breast Cancer: Targets and Therapy 2014:6 179–189
- 9) Ibrahim T; Larsen S; Hashish S, Harling H. Metronomic Chemotherapy for Pre-Treated Metastatic Pancreatic Cancer. Br J Cancer Res 2019;3: 286 91
- 10) Lundberg HE, Holand T, Holo H, Larsen S. Increased serum osteocalcin levels and vitamin K status by daily cheese intake. Int J Clin Trials. 2020 May;7(2):55-65.

### **B**: Lecturing experience

- 1) Every year since 1987, I have lectured PhD/DSc candidates in "Controlled clinical research methodology"; "Medical Statistics" and "Scientific writing"
- 2) Written 9 compendiums in these three fields
- 3) Arranged and headed 12 seminars in medical science

### C: Distinction

| • | Astra Meditec research Award | 1991 |
|---|------------------------------|-------------|
| • | Glaxo Research Award | 1994 |
| • | IEA/JOSE_ Best Paper Award | 2003 – 2005 |
| • | Pegasus research Award | 2005 |
| • | Norecopas 3R-Award | 2015 |

### D: Memberships

| • | Norwegian Statistical Society | Since 1975 |
|---|-------------------------------------------------|------------|
| • | Norwegian Society | Since 1979 |
| • | International Society of Clinical Biostatistics | Since 1984 |
| • | American Society of Clinical Oncology (ASCO) | Since 2000 |

### E: First publication in different field

- Design of Controlled Clinical Trial (first publication 1979)
- Clinical Trial Methodology (first publication 1978)
- Medical Statistics
  - o Estimation and predication (first publication 1978)
  - Discriminate analysis (first publication 1985)
  - o Sequential Analysis (first publication 1987)
  - Maximum probability estimation (first publication 1978)

| Signature: | | initials: SEL |
|-------------------------|----------------|---------------|
| Date prepared: February | <i>y</i> 2021. | |

BulbiCam; Validity study: